

#### **CLINICAL STUDY PROTOCOL**

TITLE: A Phase II, Randomized, Double-Blind, Vehicle Controlled Study

of the Efficacy, Safety, and Tolerability of B244 Topical Spray for

the Treatment of Pruritus in Adults with a History of Atopic

Dermatitis

IND Number: 17485

Protocol Number: PRB244-01

Protocol Version/Date: Amendment 3 / 28-FEB-2020

Development Phase: Phase 2

Sponsor: AOBiome Therapeutics

125 Cambridgepark Drive Cambridge, MA 02140

USA

Any and all information presented in this document shall be treated as confidential and shall remain the exclusive property of AOBiome Therapeutics (or any of its affiliated companies). The use of such confidential information must be restricted to the recipient for the agreed purpose and must not be disclosed, published or otherwise communicated to any unauthorized persons, for any reasons, in any form whatsoever without the prior written consent of AOBiome Therapeutics (or the concerned affiliated company).

# **Revision Chronology**

| Original | September 25, 2019 |
|-------------|--------------------|
| Amendment 1 | November 07, 2019 |
| Amendment 2 | January 06, 2020 |
| Amendment 3 | February 28, 2020 |

# SIGNATURE PAGE FOR INVESTIGATOR(S)

| TITLE: | A Phase II, Randomized, Double-Blind, Vehicle Controlled Study of the Efficacy, Safety, and Tolerability of B244 Topical Spray for the Treatment of Pruritus in Adults with a History of Atopic Dermatitis |
|---|---|
| IND Number: | 17485 |
| Protocol Number: | PRB244-01 |
| Protocol Version/Date: | Amendment 3 / 28-FEB-2020 |
| Development Phase: | Phase 2 |
| Sponsor: | AOBiome Therapeutics<br>125 Cambridgepark Drive<br>Cambridge, MA 02140<br>USA |
| I have read the protocol and agree to conduct this study in accordance with the protocol, all relevant laws and regulations in force at the time, International Conference on Harmonisation Guidelines for Good Clinical Practices, and the Declaration of Helsinki. | |
| Principal Investigator's printed name | |
| Principal Investigator's signa | ture Date (DD-MMM-YYYY) |

# SPONSOR PROTOCOL APPROVAL SIGNATURE(S)

| TITLE: | A Phase II, Randomized, Double-Bli<br>of the Efficacy, Safety, and Tolerabil<br>the Treatment of Pruritus in Adults w<br>Dermatitis | ity of B244 Topical Spray for |
|---|---|---|
| IND Number: | 17485 | |
| Protocol Number: | PRB244-01 | |
| Protocol Version/Date: | Amendment 3 / 28-FEB-2020 | |
| Development Phase: | Phase 2 | |
| Sponsor: | AOBiome Therapeutics<br>125 Cambridgepark Drive<br>Cambridge, MA 02140<br>USA | |
| relevant laws and regulations | agree to conduct this study in accordant in force at the time, International Con Practices, and the Declaration of Hels | ference on Harmonisation |
| Approved by: | | |
| 7400 L | | 28-Feb-2020 |
| Hyun Kim, Ph.D. | | Date (DD-MMM-YYYY) |
| Head of Clinical Operations | | |
| 11 ( ) | | |
| M | D | 28-Feb-2020 |
| Judith Ng-Cashin, M.D. | | Date (DD-MMM-YYYY) |
| Chief Medical Officer | | |

Protocol PRB244-01

Amendment 3 28-FEB-2020

## PROTOCOL SYNOPSIS

| Title | A Phase II, Randomized, Double-Blind, Vehicle Controlled Study of the Efficacy, Safety, and Tolerability of B244 Topical Spray for the Treatment of Pruritus in Adults with a History of Atopic Dermatitis |
|---|---|
| Protocol Number | PRB244-01 |
| Sponsor | AOBiome Therapeutics |
| Development Phase | II |
| Study Objectives | Primary objective: • To assess the efficacy of B244 in the treatment of pruritus in adults with a history of atopic dermatitis. |
| | <ul> <li>Secondary objectives:</li> <li>To assess the safety and tolerability of B244 in adults with a history of atopic dermatitis.</li> </ul> |
| Study Design | This is a double-blind, randomized, vehicle-controlled study to assess the efficacy, safety, and tolerability of 2 doses of B244 for the treatment of pruritus in adults with a history of atopic dermatitis. Subjects who meet the study entry criteria will be randomized in a 1:1:1 ratio to receive twice daily topical doses of B244 at 1x10 <sup>10</sup> cells/ml (O.D. 5.0), 4 x10 <sup>10</sup> cells/ml (O.D. 20.0) or vehicle (control) for 4 weeks. The total duration of the study will be approximately 11 weeks. The study will be conducted at approximately 50 study sites. |
| | At Screening and Baseline, all subjects must have atopic dermatitis, which involves a minimum of 10% and a maximum of 40% body surface area, score of $\geq$ 7 points on the NRS scale and static IGA of 2-3. |
| | The total duration of the study will be approximately 11 weeks. Participants will report for a Screening visit and if all inclusion/exclusion criteria are met, subjects will go through a two-week washout phase before reporting for a Baseline visit. At the baseline visit, eligible subjects will be randomly assigned to receive B244 1x10 <sup>10</sup> cells/ml, B244 4x10 <sup>10</sup> cells/ml or vehicle. Subjects will come in for Week 2 and Week 4 visits. After completion of the 4-week treatment period, all subjects will enter a 4-week follow-up period. Participants |

| | who have discontinued the study early will be evaluated by the Investigator at |
|---|---|
| | the Early Termination Visit within 7 days after their last dose of study drug. |
| | The primary efficacy endpoint will be assessed after Week 4 of treatment. |
| Number of patients planned for randomization | Approximately 576 subjects (192 per treatment group) will be enrolled and randomized in the study. |
| Study Population | Male and female adults 18 to 65 years of age with pruritus and a history of atopic dermatitis. |
| Inclusion Criteria: | |
| | 1. Male and female subjects 18 to 65 years of age. |
| | 2. Pruritus of at least 4 weeks duration prior to the initial Screening visit and during the 2 week washout period. |
| | <ul> <li>a. Subjects using stable doses of oral H1 antihistamines at the initial Screening visit must be willing to continue these at the same doses and frequencies throughout the study inclusive of the follow-up period.</li> <li>3. Worst Itch Numeric Rating Scale (WI-NRS) score ≥ 7 in the 24-hour period prior to the initial Screening as well as Baseline visits.</li> <li>4. Average weekly WI-NRS score ≥6 for each week of the washout period, as recorded in the eDiary.</li> <li>5. A history of atopic dermatitis for greater than 12 months consistent with a diagnosis of atopic dermatitis, as defined by the 2014 American Academy of Dermatology (AAD) Guidelines of Care for the</li> </ul> |
| | Management of Atopic Dermatitis. <sup>1</sup> a. Subjects using bland emollients at the initial Screening visit will be allowed to continue to use their emollient of choice at the same dose and frequency throughout the study. b. Subjects using low- to mid-potency topical corticosteroids at the initial Screening visit will be allowed to use their topical corticosteroid of choice at the same dose and frequency no more than 7 days per month throughout the study as rescue medication. 6. A minimum of 10% and not more than 40% of the subjects' BSA affected by atopic dermatitis (affected is defined by physical examination findings: erythema, edema, scaling, lichenification, |

excoriation, with the excoriation serving as the physical examination correlate of pruritus) at Screening and Baseline.

- a. Subjects' BSA can include face and body OR body alone BUT NOT face alone.
- 7. An Investigator Global Assessment (IGA) score of 2-3 at Screening and Baseline.
- 8. Willing and able to complete once-daily eDiary entries within a consistent timeframe for the duration of the study and have ≥80% eDiary compliance rate during the washout period.
- 9. Judged to be in good health in the investigator's opinion.

#### **Exclusion Criteria:**

- 1. Clearly defined etiology for pruritus other than atopic dermatitis. These include but are not limited to urticaria, psoriasis or other non-atopic dermatologic conditions, hepatic or renal disease, psychogenic pruritus, drug reaction, untreated hyperthyroidism, parasite presence and presence of acute infection either systemically or in the AD lesions.
- 2. Presence of any acute condition which may risk inducing an atopic dermatitis flare during the course of the study, such as impetigo or active herpes simplex infection.
- 3. Treatment with systemic corticosteroids within 4 weeks prior to randomization.
- 4. Treatment with Class III or higher potency topical corticosteroids or any topical anti-pruritic therapies (other than stable doses of low- or mid-potency topical corticosteroids or bland emollients) within 4 weeks prior to randomization.
- 5. Treatment with systemic therapies with recognized anti-pruritic (e.g. tricyclic antidepressants, sedatives, tranquilizers, gabapentin, marijuana or other cannabinoids, opioid receptor agonists/antagonists) or pruritic (e.g. opioids, angiotensin-converting enzyme inhibitors, cocaine, antimalarials) properties within 4 weeks prior to randomization.
  - a. Stable doses of H1 antihistamines will be permitted. Subjects must be willing to continue these at the same doses and frequencies throughout the study inclusive of the follow-up period.
- 6. Any clinically significant changes in type, dose, or frequency of bland emollients, low- or mid-potency corticosteroids, and/or oral H1 antihistamines throughout the study from screening to follow-up.
- 7. Treatment with systemic immunosuppressive/ immunomodulatory therapies within 4 weeks prior to randomization (including but not

| | <ul> <li>limited to phosphodiesterase-4 inhibitors, cyclosporine, mycophenolate-mofetil, methotrexate, azathioprine, interferon-gamma, or phototherapy).</li> <li>8. Treatment with biologic therapies within 12 weeks or 5 half-lives prior to randomization, whichever is longer.</li> <li>9. Use of an indoor tanning facility within 4 weeks prior to randomization.</li> <li>10. Treatment with any investigational therapy within 4 weeks prior to randomization.</li> <li>11. Allergen immunotherapy within 6 months prior to randomization.</li> <li>12. Prior use of AO+ Mist.</li> <li>13. History of malignancy within 5 years prior to randomization, with the exception of completely treated and non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin.</li> </ul> |
|---|---|
| | <ul> <li>14. History of a major psychiatric condition (including major depressive disorder, bipolar disorder, or schizophrenia), suicidal ideation, or suicide attempt.</li> <li>15. Known active hepatitis infection.</li> <li>16. Known history of human immunodeficiency virus (HIV) infection.</li> <li>17. Presence of any medical condition or disability that, in the investigator's opinion, could interfere with the assessment of safety or efficacy in this trial or compromise the safety of the subject.</li> <li>18. Currently pregnant or breastfeeding, or male subject with a pregnant or breastfeeding partner.</li> <li>19. Females of childbearing potential who are unable or unwilling to practice highly effective contraception (pregnancy prevention); fertile males who are unable or unwilling to use condoms with female partners of childbearing potential.</li> </ul> |
| Study Drug | 1) B244 1x10 <sup>10</sup> cells/ml (O.D. 5.0)<br>2) B244 4x10 <sup>10</sup> cells/ml (O.D. 20.0)<br>3) Vehicle |
| Dose Regimen | Subjects will apply 10 pumps of IP per application to all affected areas twice-a-day (i.e. 10 pumps in the morning and 10 pumps again at night) for 4 Weeks. |
| Efficacy Endpoints | The key primary efficacy endpoint is as follows: • Mean change in WI-NRS from baseline to Week 4 |

| | <ul> <li>Additional secondary efficacy endpoints include the following: <ul> <li>Proportion of subjects with ≥4 point improvement in WI-NRS from baseline to Week 4</li> <li>Proportion of subjects with any improvement in WI-NRS from baseline to Week 4</li> <li>Mean change in AI-NRS from baseline to Week 4</li> <li>Proportion of subjects with ≥4 point improvement in AI-NRS from baseline to Week 4</li> <li>Proportion of subjects with any improvement in AI-NRS from baseline to Week 4</li> <li>Mean change in WI-NRS from baseline to Week 2</li> <li>Proportion of subjects with ≥4 point improvement in WI-NRS from baseline to Week 2</li> </ul> </li> </ul> |
|---|---|
| | <ul> <li>Mean change in POEM from baseline to Week 4</li> </ul> |
| | <ul> <li>Mean change in 5-D Pruritus Scale from baseline to Week 4</li> </ul> |
| | Exploratory endpoints include the following: |
| | Mean change in IGA from baseline to Week 4 |
| | Mean change in EASI from baseline to Week 4 |
| Safety Endpoints | Safety and tolerability endpoints include the following: |
| | Incidence of treatment-emergent adverse events (TEAEs) and serious |
| | adverse events (SAEs) |
| | Changes in vital signs and clinical laboratory parameters following |
| | study drug exposure |
| | Changes in local skin tolerability following application of study drug |
| Assessment Schedule: | All subjects will attend a screening visit not more than 21 days prior to |
| | Baseline (Day 0). Subjects will be required to return to the clinic at Baseline, |
| | Day 14 (Week 2) and Day 28 (Week 4). All subjects will be asked to attend a |
| | Week 8 follow-up visit 4 weeks (28 days (±3) days) after the last dose of study |
| | medication. |
| Statistical Considerations: | Sample Size: |
| | Approximately 576 subjects may be enrolled to account for 16.7% drop out rate prior to completing the study. |
| | A total of 160 evaluable subjects per group (480 total) are required to achieve |
| | at least 80% to detect a pairwise difference of 0.65 in mean WI-NRS change |
| | from baseline to Week 4 between one of two active doses of B244 and vehicle |
| | control when assuming a standard deviation of 2.5 and applying a Dunnett |

Testing Method at a one-sided familywise error rate of 0.10.

### **Populations:**

- ITT population: All subjects who are enrolled and apply at least 1 dose of study treatment will be included in the Intent to Treat (ITT) population. The ITT population will be the primary population for safety and efficacy assessments.
- Per Protocol (PP) population: All subjects in the ITT population without any protocol deviations that may have an impact on the efficacy assessments, who complete their Week 4 visit, and who administer at least 50% of investigational product (IP), will be included in the Per Protocol (PP) population.
- Safety Population: All subjects treated with at least one dose of IP.

#### Efficacy Analysis:

Efficacy analysis will be performed on the ITT population with some supportive analysis on the PP population. Regression models will include all eligible subjects for the respective analysis, from the 3 treatment arms.

Hypothesis tests for the primary efficacy endpoint will be performed using a Dunnett Testing Method, applying pairwise comparisons of each respective B244 dose group to vehicle using a one-sided familywise error rate of 0.10. No additional adjustments will be made for multiple testing.

Additional supportive analyses may be performed combining the B244 dose groups in comparison against vehicle and comparison of the B244 groups to one another.

The frequency and rate of NRS responders at Week 4 (≥4 point change from baseline in NRS) will be reported and compared between treatment groups using a logistic regression model.

Continuous measures of change from baseline to Week 1, Week 2, Week 3, Week 4, Week 8 for AI-NRS and WI-NRS; and change from baseline to Week 2, Week 4, Week 8 for POEM and 5-D Pruritus Scale will be analyzed using mixed models with repeated measures (MMRM) to account for within-subject variability over time. Comparisons at each time point will be performed within the longitudinal model.

#### Safety Analysis:

| | Analysis of safety measures will be performed on the Safety Population, including all treated subjects. |
|---|---|
| | The incidence of all adverse events (AEs) and treatment-related AEs will be tabulated by treatment received. These AEs will be classified by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). The incidence and severity of changes in local tolerability and adverse reactions will be collected as a solicited AE of special interest. |
| | For incidence reporting, if a subject reported more than one AE that was coded to the same system organ class or preferred term, the subject will be counted only once for that specific system organ class or preferred term. An overview of AEs, which includes subject incidence of AEs, treatment-related AEs, AEs by severity, SAEs, deaths, and AEs leading to discontinuation, will be presented. |
| | Summaries of IP exposure, clinical laboratory measures, vital signs, rescue medications, and concomitant medications will be presented. |
| Study Sites | Approximately 50 study sites |
| Expected Duration of Subject's Participation | Approximately 11 weeks: Up to 3 weeks of screening, 4 weeks of treatment, and a follow-up period of 4 weeks. |

This study will be conducted in accordance with the Guidelines of Good Clinical Practices (GCPs).

## **Table of Contents**

| 1 S | STUDY SCHEMA | |
|---|---|---|
| 2 I | INTRODUCTION | |
| 2.1 | Background | 18 |
| 2.2 | Clinical Experience | 18 |
| 2.3 | Safety Profile | 20 |
| 2.4 | Rationale for the Study | 20 |
| 3 S | STUDY OBJECTIVES | |
| 3.1 | Primary Objective | 21 |
| 3.2 | Secondary Objectives | 21 |
| 4 E | ENDPOINTS | |
| 4.1 | Efficacy | 21 |
| 4.2 | Safety & Tolerability | 22 |
| 5 S | STUDY DESIGN | 22 |
| 6 S | SELECTION OF STUDY PARTICIPANTS | 23 |
| 6.1 | Number of Participants Planned | 23 |
| 6.2 | Inclusion Criteria | 23 |
| 6.3 | Exclusion Criteria | 23 |
| 7 F | PARTICIPANT ENROLLMENT | |
| 7.1 | Consenting Participants | 25 |
| 7.2 | Screening for Eligibility | 25 |
| 7.3 | Study Withdrawal and Withdrawal from Investigational Product 25 | and Stopping Criteria |
| 7.4 | Early Termination | 26 |
| <b>7.5</b> | Lifestyle Considerations | <b>27</b> |
| 8 S | STUDY TREATMENT | |
| 8.1 | Investigational Product | 27 |
| 8.2 | Dose Changes | 28 |
| 8.3 | Storage conditions | 28 |
| 8.4 | Description of Blinding Method | 29 |

| 8.5 | Treatment Assignments: | 29 |
|---|---|---|
| 8.6 | Treatment Compliance | 29 |
| 8.7 | Treatment Application | 30 |
| 8.8 | Treatment of Investigational Product Overdose | 31 |
| 8.9 | Study Drug Discontinuation | 31 |
| 8.10 | Product Accountability | 32 |
| 8.11 | Unblinding Procedures | |
| 8.12 | Retrieval and Destruction of Investigational Product | |
| 8.13 | Concomitant and Excluded Therapies | |
| 8.13. | | |
| 8.13. | | |
| 8.14 | Rescue Medications | 34 |
| 8.14. | | |
| 8.14. | | |
| 8.15 | Handling of Investigational Product | 36 |
| 9 CO | NTRACEPTION REQUIREMENTS | 36 |
| 10 S | TUDY PROCEDURES | 37 |
| 10.1 | Pre-screening procedures | |
| 10.2 | Informed Consent Procedures | |
| 10.3 | Study Assessments | |
| 10.4 | Inclusion procedures | |
| 10.5 | Timing of patient's visits to the clinic | |
| <b>10.6</b><br>10.6. | Description by type of visit | |
| 10.6. | <b>c</b> | |
| 10.6. | | |
| 10.6. | 4 Day 5- Phone call to patient | 39 |
| 10.6. | 2 2 3 1 : with 2 3 2 0 00 may 1 10 100 | |
| 10.6. | · J · | |
| 10.6. | $\mathbf{I}$ | |
| 10.6. | 8 Early Termination Visit | 41 |
| 11 S | TUDY ASSESSMENTS | 41 |
| 11.1.1 | Vital Signs | 41 |
| 11.1.2 | Physical Examinations | 41 |
| 11.1.3 | Laboratory Assessments | 42 |
| 11.2 | Efficacy Assessments | 42 |
| 11.2. | · | |
| 11.2.3 | Itch Numeric Rating Scale | 43 |
| Protocol Pl | 9 | |

| 11.2 | 2.4 Investigator Global Assessment Score (IGA) | 44 |
|---|---|---|
| 11.2 | 2.5 5-D Pruritus Scale | 44 |
| 11.3 | 8 eDiary and Efficacy Assessments | 44 |
| 11.4 | Patient Reported Local Tolerability | 45 |
| 11.5 | 5 Pregnancy Reporting | 45 |
| 11.6 | Study Completion | 45 |
| 11.7 | Subject Withdrawal Criteria | 45 |
| 12 | STATISTICAL CONSIDERATIONS | 46 |
| 12.1 | Sample Size | 46 |
| 12.2 | Populations for Analysis | 46 |
| 12.3 | B Data Analysis | 46 |
| | 2.3.1 Disposition | |
| 12.4 | | |
| | 2.4.1 Definitions | |
| | 2.4.2 Adverse Events | |
| | <ul><li>2.4.3 Deaths and Serious Adverse Events.</li><li>2.4.4 Adverse Events leading to treatment discontinuation.</li></ul> | |
| 12.5 | - | |
| 12.6 | • | |
| 12.7 | | |
| 13 | ADVERSE EVENTS (AE) AND SERIOUS ADVERSE EVENTS (SAE) | |
| 13.1 | | |
| 13.2 | Definition of a SAE | 49 |
| 13.3 | Time-period, Frequency, and Method of Detecting AEs and SAEs | 50 |
| 13.4 | | |
| 13.5 | 5 Evaluating AEs and SAEs | 51 |
| 1 | 3.5.1 Severity Rating | 51 |
| | 3.5.2 Relationship to Investigational product (IP) | |
| 13.6 | • | |
| 13.7 | | |
| 14 | ETHICAL AND REGULATORY STANDARDS | 53 |
| 14.1 | Ethical Conduct of Study | 53 |
| 14.2 | 2 Laws and Regulations | 54 |
| 14.3 | Informed Consent | 54 |
| 14.4 | Institutional Review Board/Independent Ethics Committee (IRB/EC) | 55 |
| Protoco | ol PRB244-01 | |

| 14.5 | Clinical Monitoring/Record Keeping | 55 |
|---|---|---|
| 15 | ADMINISTRATIVE RULES | 56 |
| 15.1 | Curriculum Vitae | 56 |
| 15.2 | Archiving of Study Documentation | 56 |
| 15.3 | Internal Safety Review Committee | 56 |
| 16 | STUDY MONITORING | 56 |
| 16.1 | Responsibilities of the Investigator(s) | 56 |
| 16.2 | Responsibilities of the Sponsor | 57 |
| 16.3 | Source document requirements | 57 |
| 16.4 | Use and completion of Case Report Forms (CRFs) and additional requests | 57 |
| <i>17</i> | PUBLICATIONS | 58 |
| 18 | PROTOCOL ADHERENCE | 59 |
| 19 | CLINICAL TRIAL PROTOCOL AMENDMENTS | 59 |
| 20 | CONFIDENTIALITY | 59 |
| 21 | PROPERTY RIGHTS | 59 |
| 22 | DATA PROTECTION | 60 |
| 23 | SPONSOR AUDITS AND INSPECTIONS BY REGULATORY AGENCIES | 60 |
| 24 | PREMATURE DISCONTINUATION OF THE STUDY OR PREMATURE CLO | SE- |
| OUT ( | OF A SITE | 61 |
| 24.1 | v 1 | |
| 24.2 | Decided by the Investigator | 61 |
| 25 | CLINICAL TRIAL PROTOCOL AMENDMENTS | 61 |
| <i>26</i> | REFERENCES | 62 |
| APPE | NDIX A: SCHEDULE OF EVENTS | 63 |
| APPE. | NDIX B: EXCLUDED MEDICATIONS/THERAPY | 68 |
| APPE | NDIX C: EASI SCORE | 70 |
| APPE | NDIX D: PATIENT ORIENTED ECZEMA MEASURE (POEM) | 78 |
| APPE | NDIX E: IGA | 80 |
| APPE | NDIX F: 5-D PRURITUS SCALE | 81 |
| APPE | NDIX G: PATIENT REPORTED LOCAL TOLERABILITY | 82 |

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| AD | Atopic Dermatitis |
|--------------------|-------------------------------------------|
| AE | Adverse Event |
| AI | Average Itch |
| AMO | Ammonia Monooxygenase |
| AOB | Ammonia Oxidizing Bacteria |
| BID | Twice-Daily |
| CRF | Case Report Form |
| EASI | Eczema Area and Severity Index |
| E/T | Early Termination |
| FDA | Food and Drug Administration |
| HAO | NH <sub>2</sub> OH oxidoreductase |
| HbsAg | Hepatitis B Virus Surface Antigen |
| HCV Ab | Hepatitis C Virus Antibody |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IGA | Investigator Global Assessment |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| NH <sub>2</sub> OH | Hydroxylamine |
| NH <sub>3</sub> | Ammonia |
| NO | Nitric oxide |
| NO <sub>2</sub> - | Nitrite |
| NRS | Itch Numeric Rating Scale |
| PCP | Primary Care Physician |
| POEM | Patient Oriented Eczema Measure |
| SAE | Serious Adverse Event |
| SPM | Study Procedures Manual |
| VAS | Visual Analog Scale |
| WI | Worst Itch |

#### 1 STUDY SCHEMA



#### 2 INTRODUCTION

#### 2.1 **Background**

Ammonia oxidizing bacteria (AOB) are essential for the initial step in environmental nitrification processes, specifically the oxidation of ammonia (NH<sub>3</sub>) to nitrite (NO<sub>2</sub>-). Nitrosomonas are Gram-negative chemolithoautotrophic betaproteobacteria that obtain energy solely from NH<sub>3</sub> oxidation, while fixing CO<sub>2</sub> for their carbon needs<sup>2</sup>. Oxidation of NH<sub>3</sub> proceeds in two steps (Figure 1) leading to sequential generation of hydroxylamine (NH<sub>2</sub>OH) and NO<sub>2</sub>- that require two enzyme complexes: the membrane-bound ammonia monooxygenase (AMO) comprised of subunits AmoA, AmoB and AmoC; and the periplasmic NH<sub>2</sub>OH oxidoreductase (HAO). In addition to high NO<sub>2</sub>- levels, NH<sub>3</sub> oxidation leads to nitric oxide (NO) and N<sub>2</sub>O production through two independent pathways downstream of NH<sub>2</sub>OH production: nitrifier denitrification and NH<sub>2</sub>OH oxidation<sup>3</sup>.

Figure 1



B244 is a purified a strain of *Nitrosomonas eutropha* originally isolated from soil samples. Sequencing of the B244 genome revealed a distinct genetic profile from that of other published Nitrosomonas strains and AOB genomes. Based on in vitro co-culture studies, B244 was able to reduce survival of pathogenic bacteria. Nitrite generation from ammonia concurrently with medium acidification by B244 led to strong antibacterial effects and a marked reduction (~100fold) in viable counts of methicillin-resistant Staphylococcus aureus and Pseudomonas aeruginosa, two pathogens frequently isolated from infected skin and wound sites. In contrast, control cultures with B244 in the absence of ammonium or with heat-killed B244 supplemented with ammonium, had no antibacterial effects. The unique metabolic and antimicrobial activity of Nitrosomonas, in combination with their lack of virulence render these bacteria as attractive candidates for topical delivery of nitrite and nitric oxide on human skin with potential to improve health in both normal and abnormal skin conditions or wound sites. NO-releasing drugs or NO donors have also shown activity against *Propionibacterium acnes* and other pathogenic bacteria, anti-inflammatory activity, and inhibition of lipogenesis by insulin-stimulated immortal sebocytes<sup>4-6</sup>.

#### 2.2 **Clinical Experience**

B244 is being developed as a 'live topical' to provide a natural source of AOB and NO/NO<sub>2</sub> to the human skin.

AOBiome's first Phase 1b/2a clinical trial titled, "A Double Blind, Vehicle-Controlled, Single Center, Randomized, Sequential, Ascending 14-Day Multiple Dose Study in Subjects with Acne Vulgaris to Evaluate the Safety, Tolerability and Preliminary Efficacy of B244 Delivered as a Topical Spray" was completed in 2016 where 36 participants with clinical diagnosis of facial acne vulgaris were randomized to receive ascending doses of investigational product (IP) over 14 days. Safety analyses have been completed and there has been no attributable drug related SAEs reported. In addition, a Phase 2b/3 clinical trial titled, "A Randomized, Double Blinded, Phase IIb/III, Decentralized Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Participants with Mild to Moderate Acne Vulgaris in 372 patients with clinical diagnosis of facial acne" has been completed. B244 was safe and well tolerated with no attributable drug related SAEs. Efficacy was supported by statistically significant 2-point reduction in IGA with B244 and a trend in the reduction of the number of inflammatory lesions compared to vehicle.

A study titled, "A Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized, Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Atopic Dermatitis" has recently been completed. A total of 122 subjects were enrolled and randomized in a 1:1 ratio to receive B244 or vehicle in the study. Overall, there were no unexpected safety signals observed following treatment with B244. A total of 30 (25%) subjects experienced at least 1 treatment-emergent adverse events (TEAE) during the study, including 16 (26%) subjects in the B244 treatment group and 14 (23%) subjects in the vehicle group.

AOBiome completed a Phase Ib study in pediatric and adolescent subjects aged 2-17 years of age. A study titled, "An Open-label, Multicenter, Phase Ib Study of B244 Delivered as a Topical Spray to Assess Safety in Pediatric Subjects aged 2 to 17 years with Atopic Dermatitis" enrolled a total of 28 subjects across 3 cohorts. Overall, there were no unexpected safety signals observed following treatment with B244 in pediatric subjects with atopic dermatitis. The B244 spray was well tolerated and not associated with any increased pain or redness at the application site.

"A Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Mild to Moderate Rosacea" has been completed with a total of 140 subjects randomized. Generally, there were no unexpected safety signals observed following treatment with B244. Overall, 31 (22.1) subjects had experienced at least one treatment emergent adverse event of which 19 (26.0%) subjects in B244 spray group and 12 (17.9%) in the Vehicle group.

In addition, other topical development programs with B244 include hypertension. A study titled, "A Prospective, Controlled, Double Blinded, Multicenter, Randomized, Vehicle Controlled, Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects with Elevated Blood Pressure" has been completed. Safety data indicated that B244 was safe and well tolerated. Overall, 16% of subjects experienced at least 1 TEAE during the study with comparable incidence in the B244 and Vehicle groups. Overall, there were no unexpected safety signals observed following treatment with B244.

Moreover, intranasal application of B244 is being developed for the treatment of allergic rhinitis and migraines. A rat toxicology study performed by intranasal administration of B244 twice daily for 28 days found that B244 was safe and well tolerated in rats at levels of up to the maximum dose 8x10<sup>9</sup> cell/mL. A study titled, "A Prospective, Controlled, Double Blinded, Single Center, Randomized, 3 arm, Phase 1b/2a Study to Assess the Safety, Tolerability, and Preliminary Efficacy of B244 Delivered as an Intranasal Spray in Healthy Volunteers and Subjects with Seasonal Allergic Rhinitis" has been completed. In addition, a study titled "A Prospective, Randomized, Vehicle-Controlled, Double-Blind, Phase 2 Study to Assess the Safety, Tolerability, and Efficacy of B244 Delivered as an Intranasal Spray for Preventive Treatment in Subjects with Episodic Migraine" is in progress.

## 2.3 Safety Profile

To date, there have been no reported infections or health risks associated with topical application or ingestion of *Nitrosomonas* species. The absence of any illnesses attributed to these bacteria despite our widespread exposure indicates that they pose a minimal health risk, if any at all. Infection or tissue damage by *Nitrosomonas* is unlikely, because the sequenced genomes of several *Nitrosomonas* and other AOB lack genes encoding cytotoxins, or other known bacterial virulence factors. Further, AOB are slow growing, as compared to most heterotrophic bacteria, with optimum doubling times of 8 hours or higher. In particular, *Nitrosomonas* growth is rate limited by the availability of ammonia requiring the oxidation of 27 moles NH<sub>3</sub>/mole CO<sub>2</sub> fixed. Due to their dependence on ammonia for their growth, the numbers of *Nitrosomonas* on the skin will be necessarily limited and naturally regulated by the amount of ammonia produced in sweat. This would ensure that the amount of nitrite and NO generated would be relatively low, without any adverse effects.

#### 2.4 Rationale for the Study

Eczema or Atopic dermatitis is an inflammatory skin condition that affects nearly 20% of children and between 2-10% of adults<sup>7</sup>. Disease prevalence has steadily grown in the last 30 years, resulting in a growing field of atopic dermatitis research<sup>8</sup>.

Pruritus is a common morbidity associated with Atopic Dermatitis, and its management remains a challenge for physicians. Pruritus is defined as an urge or unpleasant sensation that produces the urge to scratch<sup>9</sup>. Modern treatment no longer consists of antihistamines alone. Anti-inflammatory, antiseptic, as well as antipruritic therapies to address the epidermal barrier as well as immunomodulation or infection are now used in clinical practice<sup>9</sup>. Mild pruritus may be controlled with topical therapies, while moderate to severe pruritus requires combination treatment, consisting of antipruritic and immunosuppressive drugs, phototherapy, and topical compounds<sup>9</sup>.

While the complete pathophysiology of pruritus remains unclear, histamines are one of the most potent mediators in AD related pruritus. The itch cycle exacerbates damage to the epidermal barrier leading to water loss and dryness, thereby creating a hospitable environment for skin Protocol PRB244-01

pathogens, which cause infections and flare up symptoms. *Staphylococcus aureus* is consistently found in eczematous skin lesions in patients with AD. Correlation between the severity of the disease and presence of *Staphylococcus aureus* has been well established and it has been shown that the presence of bacteria is an important factor in skin aggravation <sup>10</sup>. The goal of therapy for AD is to restore the epidermal barrier function and reduce skin inflammation, thereby alleviating symptoms and intensity of AD associated pruritus. However, systemic antibiotic use is controversial.

B244 has been developed as a topical application of a natural source of AOB and NO/NOx to the human skin. We hypothesize that application of AOB to eczematous skin may reduce *Staphylococcus aureus* skin load and normalize the inflammatory response by reducing Th2 activation.

The primary purpose of this study is to evaluate the efficacy and safety of B244 in the treatment of pruritus in adults with a history of atopic dermatitis.

#### 3 STUDY OBJECTIVES

#### 3.1 Primary Objective

• To assess the efficacy of B244 in the treatment of pruritus in adults with a history of atopic dermatitis.

#### 3.2 Secondary Objectives

• To assess the safety and tolerability of B244 in adults with a history of atopic dermatitis.

#### 4 ENDPOINTS

#### 4.1 Efficacy

#### 4.1.1 Primary

• Mean change in WI-NRS from baseline to Week 4

#### 4.1.2 Secondary

- Proportion of patients with ≥4 point improvement in WI-NRS from baseline to Week 4
- Proportion of subjects with any improvement in WI-NRS from baseline to Week 4
- Mean change in AI-NRS from baseline to Week 4
- Proportion of subjects with  $\geq 4$  point improvement in AI-NRS from baseline to Week 4
- Proportion of subjects with any improvement in AI-NRS from baseline to Week 4
- Mean change in WI-NRS from baseline to Week 2
- Proportion of subjects with ≥4 point improvement in WI-NRS from baseline to Week 2
- Mean change in POEM from baseline to Week 4
- Mean change in 5-D Pruritus Scale from baseline to Week 4

#### 4.1.3 Exploratory

- Mean change in IGA from baseline to Week 4
- Mean change in EASI from baseline to Week 4

#### 4.2 Safety & Tolerability

Safety and tolerability endpoints include the following:

- Incidence of TEAEs and SAEs
- Changes in vital signs and clinical laboratory parameters following study drug exposure
- Changes in local skin tolerability following application of study drug

#### 5 STUDY DESIGN

- This is a Prospective, Vehicle Controlled, Double-Blind, Multicenter, Randomized Phase II Trial, comparing the effect of twice daily B244 applications for 4 weeks vs vehicle applications on treatment of mild to moderate pruritus associated with atopic dermatitis.
- Approximately 576 subjects may be enrolled.
- The total duration of the study will be approximately 11 weeks. Participants will report for a Screening visit and if all inclusion/exclusion criteria are met, subjects will go through a two-week washout phase (see Section 10.6.2) before reporting for a Baseline visit.
- After screening and baseline, participants will be randomized to one of two doses of B244 or vehicle application for 4 weeks.
- Randomization will be 1:1:1 so that an equal number of patients will be treated in each Arm of the study.
- All B244 randomized subjects will be treated at the dose of  $1x10^{10}$  cells/ml (O.D. 5.0) or  $4x10^{10}$  cells/ml (O.D. 20.0).
- Subjects must be willing and able to complete diary within a consistent time frame on a daily basis and to comply with restrictions on allowable therapies for the duration of the study.
- All subjects will attend a screening visit not more than 21 days prior to Baseline (Day 0). Subjects will be required to return to the clinic at Baseline, Day 14 (Week 2) and Day 28 (Week 4) visits. All subjects will be asked to attend a Week 8 follow-up visit 4 weeks (28 (±3) days) after the last dose of study medication.
- Subjects will apply a total of 10 pumps of IP per application across all affected areas twice-a-day (i.e. 10 pumps in the morning and 10 pumps again at night) for 4 weeks.
- Safety evaluations will consist of review of participant's medical history at screening and on-going assessment of adverse events reported throughout the study duration.

#### 6 SELECTION OF STUDY PARTICIPANTS

#### **6.1** Number of Participants Planned

Approximately 576 subjects (192 per treatment group) with pruritus and a history of atopic dermatitis will be randomized into this study.

#### 6.2 Inclusion Criteria

Deviations from inclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or participant safety. Therefore, adherence to the criteria as specified in the protocol is essential.

Participants eligible for enrollment in the study must meet all the following criteria:

- 1. Male and female subjects 18 to 65 years of age.
- 2. Pruritus of at least 4 weeks duration prior to the initial Screening visit and during the 2 week washout period.
  - a. Subjects using stable doses of oral H1 antihistamines at the initial Screening visit must be willing to continue these at the same doses and frequencies throughout the study inclusive of the follow-up period.
- 3. Worst Itch Numeric Rating Scale (WI-NRS) score  $\geq 7$  in the 24-hour period prior to the initial Screening as well as Baseline visits.
- 4. Average weekly WI-NRS score ≥6 for each week of the washout period, as recorded in the eDiary.
- 5. A history of atopic dermatitis for greater than 12 months consistent with a diagnosis of atopic dermatitis, as defined by the 2014 American Academy of Dermatology (AAD) Guidelines of Care for the Management of Atopic Dermatitis<sup>1</sup>.
  - a. Subjects using bland emollients at the initial Screening visit will be allowed to continue to use their emollient of choice at a similar dose and frequency throughout the study, if used.
  - b. Subjects using low- to mid-potency topical corticosteroids at the initial Screening visit will be allowed to use their topical corticosteroid of choice at the same dose and frequency no more than 7 days per month throughout the study as rescue medication.
- 6. A minimum of 10% and not more than 40% of the subjects' BSA affected by atopic dermatitis (*affected* is defined by physical examination findings: erythema, edema, scaling, lichenification, excoriation, with the excoriation serving as the physical examination correlate of pruritus) at Screening and Baseline.
  - a. Subjects' BSA can include face and body OR body alone BUT NOT face alone.
- 7. An Investigator Global Assessment (IGA) score of 2-3 at Screening and Baseline.
- 8. Willing and able to complete once-daily eDiary entries within a consistent timeframe for the duration of the study and have ≥80% eDiary compliance rate during the washout period.
- 9. Judged to be in good health in the investigator's opinion.

#### 6.3 Exclusion Criteria

Deviations from exclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or participant safety. Therefore, adherence to the criteria as specified in the protocol is essential.

Participants will be excluded from the study if any of the following criteria are met:

- 1. Clearly defined etiology for pruritus other than atopic dermatitis. These include but are not limited to urticaria, psoriasis or other non-atopic dermatologic conditions, hepatic or renal disease, psychogenic pruritus, drug reaction, untreated hyperthyroidism, parasite presence and presence of acute infection either systemically or in the AD lesions.
- 2. Presence of any acute condition which may risk inducing an atopic dermatitis flare during the course of the study, such as impetigo or active herpes simplex infection.
- 3. Treatment with systemic corticosteroids within 4 weeks prior to randomization.
- 4. Treatment with Class III or higher potency topical corticosteroids or any topical antipruritic therapies (other than stable doses of low- or mid-potency topical corticosteroids or bland emollients) within 4 weeks prior to randomization.
- 5. Treatment with systemic therapies with recognized anti-pruritic (e.g. tricyclic antidepressants, sedatives, tranquilizers, gabapentin, marijuana or other cannabinoids, opioid receptor agonists/antagonists) or pruritic (e.g. opioids, angiotensin-converting enzyme inhibitors, cocaine, antimalarials) properties within 4 weeks prior to randomization.
  - a. Stable doses of H1 antihistamines will be permitted. Subjects must be willing to continue these at the same doses and frequencies throughout the study inclusive of the follow-up period.
- 6. Any clinically significant changes in type, dose, or frequency of bland emollients, low- or mid-potency corticosteroids, and/or oral H1 antihistamines throughout the study from screening to follow-up.
- 7. Treatment with systemic immunosuppressive/ immunomodulatory therapies within 4 weeks prior to randomization (including but not limited to phosphodiesterase-4 inhibitors, cyclosporine, mycophenolate-mofetil, methotrexate, azathioprine, interferongamma, or phototherapy).
- 8. Treatment with biologic therapies within 12 weeks or 5 half-lives prior to randomization, whichever is longer.
- 9. Use of an indoor tanning facility within 4 weeks prior to randomization.
- 10. Treatment with any investigational therapy within 4 weeks prior to randomization.
- 11. Allergen immunotherapy within 6 months prior to randomization.
- 12. Prior use of AO+ Mist.
- 13. History of malignancy within 5 years prior to randomization, with the exception of completely treated and non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin.
- 14. History of a major psychiatric condition (including major depressive disorder, bipolar disorder, or schizophrenia), suicidal ideation, or suicide attempt.
- 15. Known active hepatitis infection.
- 16. Known history of human immunodeficiency virus (HIV) infection.

- 17. Presence of any medical condition or disability that, in the investigator's opinion, could interfere with the assessment of safety or efficacy in this trial or compromise the safety of the subject.
- 18. Currently pregnant or breastfeeding, or male subject with a pregnant or breastfeeding partner.
- 19. Females of childbearing potential who are unable or unwilling to practice highly effective contraception (pregnancy prevention); fertile males who are unable or unwilling to use condoms with female partners of childbearing potential.

#### 7 PARTICIPANT ENROLLMENT

#### 7.1 Consenting Participants

Informed consent for participation in the study must be obtained before performing any study-specific procedures.

Informed Consent Forms for enrolled participants and for participants who are not subsequently enrolled will be maintained at the study site in secure study files. Consent will be obtained by trained research study staff trained in taking informed consent. The study will be explained with the opportunity for the participant to ask questions. If a participant wishes to enter the study, a consent form will be completed and signed.

### 7.2 Screening for Eligibility

After informed consent has been obtained, to determine participant eligibility for enrollment in the study, screening assessments will be performed within 1 week (-21 to -14 days) prior to starting the Washout period (-14 to -1). All screening evaluations must be completed and reviewed to confirm that participants meet all eligibility criteria before Washout period and subsequent randomization on Day 0. Subjects will be asked to undergo a 2 week (-14 to -1) washout period prior to the Baseline procedure. During the screening, washout, treatment and follow-up periods, subjects will be asked to stop utilizing bleach or vinegar as a pruritus or atopic dermatitis therapy, as well as any other treatments described in the exclusion criteria and the Excluded Medications/Therapy (Appendix B).

All screening assessments are listed in the Time and Events Table (Appendix A). A participant must meet all inclusion criteria, and none of the exclusion criteria, to be enrolled and randomized in this study. The Investigator and team will maintain a screening log to record details of all persons screened and to confirm eligibility or record reasons for screening failure, as applicable.

# 7.3 Study Withdrawal and Withdrawal from Investigational Product and Stopping Criteria

A participant may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the Investigator.

Reasons for withdrawal (participants who refuse to complete any remaining study visits) or discontinuation (participants who prematurely stop the application) at any time during the study may include, but are not limited, to the following:

- For safety reasons, either at the discretion of the Investigator or at the participant's request
- For protocol violations at the discretion of AOBiome
- Withdrawal of consent by the Subject
- Lost to follow-up
- Due to use of concomitant therapy that could interfere with the results of the study (the Investigator will report all such information through the CRF and decide, in accordance with AOBiome, whether the participant is to be withdrawn).

The reason for participant study withdrawal will be recorded in the electronic Case Report Form (eCRF). Data from participants withdrawing from the study will be considered evaluable up to the point at which they are withdrawn using the same criteria for evaluability as for participants who complete the study.

Study stopping rules will be implemented to stop the study for safety review in the event that:

- 1 subject reports death, or
- >2 subjects report an SAE, or
- >4 subjects experience grade 3 AEs of a similar type, or
- >6 subjects experience grade 2 AEs of a similar type

when the reported SAEs or AEs are considered possibly, probably, definitely or related to the investigational product.

Atopic Dermatitis is an active disease with known seasonal and personal histories of flares and exacerbations of the patient's underlying disease state. This includes personal histories of worsening itch and itch-scratch cycles, which can lead to localized infection and localized cellulitis. A subject's known and collected clinical history should be considered by the principal investigator when determining relationship of event to the investigational product.

#### 7.4 Early Termination

Early termination from the study may occur due to loss to follow-up or withdrawal of consent by the subject. Participants who have discontinued the study early will be evaluated by the Investigator at the Early Termination Visit. See the list of assessments to be performed at the Early Termination Visit in the Time and Events Table (Appendix A). Participants with ongoing AEs or SAEs believed to be possibly related to investigational product (IP) will continue to be followed until resolution or for 30 days as warranted by the nature of the AE.

### 7.5 Lifestyle Considerations

There are no dietary or activity related restrictions for this study.

#### 7.5.1 Use of Bland Emollients During the Study

Subjects will be allowed to use their usual choice of bland emollients (e.g., lotion, moisturizer) from screening to follow-up, on an as needed basis, using specific time of use guidelines in relation to study medication application. Subjects will be allowed to use their emollient of choice at a similar dose and frequency throughout the study if used. Any clinically significant changes in type, dose, or frequency of bland emollients will not be allowed during the study. A detailed guideline will be shared with the sites and subjects to ensure consistency in study medication treatment application and relation to body washing, emollient use, and other chemical exposure to skin.

Subjects will be encouraged not to use sunscreen on the treated lesions during participation in the study. Sunscreen should be used minimally or used sparingly while in the active treatment phase (Baseline to Week 4) of the study. Alternatively, sunscreen should be washed off prior to study medication use.

Subjects who do not have atopic dermatitis on their face may apply makeup as needed. However, those subjects who have atopic dermatitis on their face and require to use makeup will be advised to use it minimally.

#### 8 STUDY TREATMENT

#### 8.1 Investigational Product

Under normal conditions of handling and administration, IP is not expected to pose significant safety risks to site staff. A Material Safety Data Sheet describing the occupational hazards and recommended handling precautions will be provided to site staff if required by local laws or will otherwise be available from the Sponsor upon request.

Investigational product must be stored in a secure area under the appropriate physical conditions for the product (2-8°C). Access to and administration of the IP will be limited to the Investigator and authorized site staff. Investigational product must be dispensed or administered only to participants enrolled in the study and in accordance with this protocol (see Section 8.6).

The Investigator is responsible for study treatment accountability, reconciliation, and record maintenance. The Investigator or designated site personnel must maintain study treatment accountability records throughout the course of the study. The responsible person(s) will document the amount of study treatment received from and returned to the sponsor and the amount administered to participants. The required accountability unit for this study will be the

bottle. Discrepancies are to be reconciled or resolved.

| Product name: | B244, 30ml/bottle | B244, 30ml/bottle | Vehicle, 30ml/bottle |
|---|---|---|---|
| Dosage form: | B244 suspension | B244 suspension | Vehicle solution |
| Unit dose strength: | 1 x 10 <sup>10</sup> cells/ml<br>(O.D. 5.0) | 4x10 <sup>10</sup> cells/ml<br>(O.D. 20.0) | 50nM Na <sub>2</sub> HPO <sub>4</sub> -<br>2mM MgCl <sub>2</sub> (pH 7.6) |
| Route/administration/duration: | Topical application<br>BID for 28 days | Topical application<br>BID for 28 days | Topical application<br>BID for 28 days |
| Dosing instructions: | Subjects will apply a total of 10 pumps of IP per application to all affected areas twice-aday (i.e., 10 pumps in the morning and 10 pumps again at night). | Subjects will apply a total of 10 pumps of IP per application to all affected areas twice-aday (i.e., 10 pumps in the morning and 10 pumps again at night). | Subjects will apply a total of 10 pumps of IP per application to all affected areas twice-aday (i.e., 10 pumps in the morning and 10 pumps again at night). |
| Physical description: | Applications should occur in the morning and at night for 4 weeks. Odorless, cloudy, | Applications should occur in the morning and at night for 4 weeks. Odorless, cloudy, | Applications should occur in the morning and at night for 4 weeks. Odorless, clear, and |
| * | light pink<br>suspension | light pink<br>suspension | colorless suspension |
| Manufacturer/source of procurement: | AOBiome, LLC | AOBiome, LLC | AOBiome, LLC |

The contents of the label will be in accordance with all applicable regulatory requirements. B244 and matching vehicle will be packaged in identical 30 ml white bottles.

## 8.2 Dose Changes

No dose changes are anticipated.

## 8.3 Storage conditions

All investigational drug supplies in the study will be stored in a secure, refrigerated (2-8°C) safe place, under the responsibility of the Investigator or other authorized individual.

#### 8.4 Description of Blinding Method

This study will be double-blinded: neither Investigator(s), nor study participants, nor those involved in the conduct of the trial (including sponsor staff) will be aware of the treatment the participants are receiving. The appearance of B244 and vehicle dispensing containers will be identical.

#### **8.5** Treatment Assignments:

This is a double-blind study. Participants will be assigned to study treatment in accordance with the randomization schedule generated for the allocation of B244 or vehicle prior to the initiation of the trial. Randomization will be centrally-based and performed using an appropriate IWRS (an automated randomization system).

Each participant scheduled to receive investigational product (IP) will receive a randomization number at the time of randomization. The randomization number will be used to identify the study medication kit assigned to the participant and indicate the treatment to be administered to that participant.

#### 8.6 Treatment Compliance

Study treatment must be dispensed or administered according to procedures described herein. Only participants enrolled in the study may receive study treatment. Only authorized site personnel may supply study treatment. Participants will record use of the study medication utilizing the study diary at the time of use each day. Participants will review study medication compliance with the Investigator or designee. Any missed doses, timing, and reason for missed dose will be recorded in the eCRF. There should be no doubling of doses to make up for missed doses. If a dose is missed, the next dose of study medication should be taken as scheduled.

Each site participating in the trial will be instructed to assess subject's compliance by weighing the investigational product at the Baseline visit, Week 2 visit, and Week 4 visit and followed every time study medication is dispensed and returned per instructions below. Sites will be provided scales, which will be calibrated prior to each use. Study personnel will be instructed to record measurements into the eCRF.

All weight measurements will be performed without the safety cap. Subjects will be dispensed 2 bottles upon randomization, and each bottle will be labeled 1 and 2 with a permanent marker at the site. Unused Bottle 1 will be vortexed, primed, and weighed without the cap by the site per treatment application instructions and dispensed to the subject who will mix and apply the first dose at the site under study staff supervision. Bottle 2 will also be vortexed, primed, and weighed at the site at the time of dispense without the cap, the cap inserted back on the bottle,

and the bottle returned to its carton unused. After the first treatment application of Bottle 1, subjects will take home both bottles where they will place Bottle 1 on the counter at room temperature for in-home application twice a day until empty. Bottle 2 will be stored in the refrigerator until Bottle 1 is empty, at which point Bottle 2 will be taken out of the refrigerator, mixed per treatment application instructions, and used. Should Bottle 1 run out during a treatment application, the subject will count the number of pumps that were made with Bottle 1 and complete the remaining number of pumps needed to achieve a total of 10 pumps using Bottle 2.

At the Week 2 visit, subjects will return any empty bottle (likely Bottle 1 since each bottle should last approximately 10 days and the subject should be on Bottle 2 at the time of visit) to the site for weight measurement (without the safety cap) to confirm usage. At this visit, a third bottle of the same treatment group will be labeled as Bottle 3 and will be vortexed, primed, and weighed at the site at the time of dispense without the cap, the cap inserted back on the bottle, and the bottle returned to its carton unused. The subject will be dispensed Bottle 3 to take home and store in the refrigerator until Bottle 2 is empty, at which point Bottle 3 is taken out of the refrigerator and used on the counter until the Week 4 visit. All empty bottles returned to the site will be collected and stored by the site in ambient temperature until return to the drug depot. If the subject is still on Bottle 1 at the Week 2 visit, the site will confirm daily dosing application and retrain the subject on the appropriate use of IP application, and the subject will continue using Bottle 1 until empty, at which point Bottle 2 is taken out of the refrigerator and used on the counter until Bottle 2 is empty, after which Bottle 3 is taken out of the refrigerator and used on the counter until the Week 4 visit. Any bottle currently in use at the time of the Week 2 visit should not be returned to the site.

At the Week 4 visit, all used and unused bottles will be returned to the site for weight measurements and storage at the site in ambient temperature until return to the drug depot.

## 8.7 Treatment Application

Subjects will receive study drug for application throughout the study. Subjects will be instructed in the use of the spray bottle and asked to self-administer the Investigational Product following a detailed instruction on treatment application that will be shared with the sites and subjects to ensure consistency in treatment application and relation to body washing, emollient use, and other chemical exposure to skin. Key guidelines include:

- The subject should wash his/her hands before applying study treatment.
- Subjects will apply a total of 10 pumps of IP per application to all affected. areas twice-aday (i.e., 10 pumps in the morning and 10 pumps again at night).
- The subject will apply the IP to the affected area twice daily (approximately 12 hours apart) for 28 consecutive days.
- Subject should mix the bottle thoroughly per instructions provided before each application and then saturate the application area well, holding the bottle approximately 6 inches away from the skin.

- Subjects will be asked to let the product air dry after each application.
- Subjects will follow instructions provided for body washing, emollient use, and other chemical exposure to skin in relation to timing of IP application.
- The spray bottle in use may be stored at ambient temperature until used up, while additional unused bottles will be stored in the refrigerator until use. DO NOT FREEZE.
- The subject will apply the IP to the worst and largest lesions first and then apply the IP to the smaller lesions. If after covering all lesions, the total number of pumps per application has not been exhausted, subject should go back and cover the worst lesions with the remaining number of pumps. However, the total number of 10 pumps allowed should not be exceeded per application.
- Subjects will be asked not to expose the treatment kit to conditions which are unnatural or harmful to the product, such as excessive heat (temperatures over 77°F [25°C] and freezing temperatures below 32°F [0°C]). Subjects may travel with their study medication but should not leave it in a hot car, outside in the cold temperatures, etc. Subjects will also be asked not to tamper or cause damage to the IP bottle.

#### 8.8 Treatment of Investigational Product Overdose

The sponsor does not recommend specific treatment for an overdose. Washing with conventional cleanser and water will remove the product. The Investigator will use clinical judgment to treat any overdose.

#### 8.9 Study Drug Discontinuation

Subjects will be discontinued from study drug treatment in the following events:

- The subject experiences a Grade 2 or higher treatment emergent AE that is assessed as likely related to study drug
- The subject receives treatment with an excluded therapy or has a clinically significant change in dose or frequency of allowed adjunctive therapies during the treatment period
- The female subject becomes pregnant or female partner of a male subject becomes pregnant or is breastfeeding

Discontinuation from study drug treatment may also occur for any of the following reasons:

- Subject decision to discontinue study drug treatment, or subject decision to withdraw consent from the study
- Any medical condition that may jeopardize the subject's safety if study drug is continued, in the investigator's and/or Sponsor's opinion
- Discontinuation is deemed to be in the best interest of the subject, in the investigator's and/or Sponsor's opinion

Subjects who discontinue treatment with study drug prior to completing the treatment period will have an ETD visit within 7 days after their last dose of study drug in addition to a follow-up visit

#### 8.10 Product Accountability

In accordance with federal and local regulatory requirements, the Investigator and designated site personnel must document the amount of investigational product dispensed to study participants, the amount returned by study participants, and amount received and returned to the sponsor, when applicable. Product accountability records must be maintained throughout the course of the trial. Any quality issue noticed with the receipt or use of an IP (deficient IP in condition, appearance, pertaining documentation, labeling, expiry date, etc.) should be promptly reported to the Sponsor, who will initiate a complaint procedure. All investigational product must be stored in a secure locked room with access limited to the Investigator and designated site personnel. Study product is to be stored in a refrigerator between 2-8°C. Maintenance of a temperature log is required. Under no circumstances will the Investigator allow IP to be used other than as directed by this Clinical Trial Protocol, or dispose of IP in any other manner.

#### **8.11 Unblinding Procedures**

The Investigator may unblind a participant's treatment assignment only in the case of emergency or in the event of a serious medical condition when knowledge of the study treatment is essential for the appropriate clinical management or welfare of the participant, as determined by the Investigator. It is preferred (but not required) that the Investigator first contacts the Medical Monitor to discuss options before unblinding the participant's treatment assignment. The Investigator must notify the Sponsor as soon as possible when a participant's treatment assignment is unblinded without revealing the treatment assignment of the unblinded participant unless that information is deemed important for the safety of participants currently in the study. The date and reason for the unblinding must be documented in the participant's study record. The Medical Monitor may unblind the treatment assignment for any participant with an SAE. If the SAE requires that an expedited regulatory report be sent to one or more regulatory agencies, a copy of the report, identifying the participant's treatment assignment, may be sent to clinical Investigators in accordance with local regulations and/or sponsor policy.

#### 8.12 Retrieval and Destruction of Investigational Product

All partially used or unused treatments will be returned to the site as brought by study participants. A detailed IP log of the returned IP shall be established.

The site will not destroy unused IP unless the Sponsor provides written authorization to the contrary. All used and unused bottles will be shipped to the authorized drug depot at the end of the study.

#### 8.13 Concomitant and Excluded Therapies

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that the subject is receiving within 30 days prior to screening and through the final study visit will be recorded on the appropriate CRF) along with:

- Reason for use.
- Dates of administration including start and end dates.
- Dosage information including dose and frequency.

Any medications started during the study (including "as needed" medications) will be recorded in the concomitant medication list as soon as the Investigational Site will become aware of the medication being added.

Details of any medication taken by the subject outside of the study center will be reviewed by the Investigator or designee on each study center visit. The Medical Monitor should be contacted if there are any questions regarding concomitant or prior therapy.

A list of excluded medications/therapy is provided in Appendix B.

Previous treatment of atopic dermatitis must be recorded irrespective of the term it was given. Acetaminophen is permitted for use any time during the study. Other concomitant medication may be considered on a case-by-case basis by the Investigator in consultation with the Medical Monitor.

Concomitant therapies include any therapies (including over-the-counter medications) used by a subject from initiation of study drug treatment through the follow-up period. A record of all medications used will be maintained for each subject throughout the study. Reported information will include a description of the type of drug, treatment period, dosing regimen, the route of administration, and drug indication.

#### **8.13.1 Permitted Medications**

Subjects using oral contraceptives, hormone-replacement therapy, or other maintenance therapies that are not Excluded Therapies (Appendix B) may continue their use during the study.

Stable doses of the following therapies for pruritus and/or atopic dermatitis will be allowed as adjunctive therapies during the study:

- Oral H1 antihistamines
- Bland emollients

A detailed guideline will be shared with the sites and subjects to ensure consistency in study medication treatment application and relation to body washing, emollient use, and other chemical exposure to skin.

Low- or mid-potency topical corticosteroids will be allowed per subjects' usual medication, frequency, and dose throughout the study from screening to washout, treatment, and follow-up periods as rescue medication up to 7 days per month.

Subjects using any of these adjunctive therapies should maintain their regimen without clinically significant changes in type, dose or frequency throughout the screening, treatment, and follow-up periods.

All participants will be screened for concomitant medications prior to inclusion into the study. Any concomitant medication to treat adverse events will be recorded in the Concomitant Medication section of the eCRF.

#### **8.13.2** Excluded Therapies

Therapies and medications that are excluded from the initial Screening visit through the follow-up period are listed in Appendix B.

#### **8.14 Rescue Medications**

#### **8.14.1** Rescue Medication Permitted During the Study

Over the course of the study, the Investigator will monitor and evaluate subject's condition and determine whether rescue therapy may be necessary. The use of medications to treat a subject's atopic dermatitis during the study will be permitted if a medical professional determines that it becomes medically necessary. Such rescue treatment should not exceed 7 days per month for the duration of the trial (screening, washout, treatment, and follow-up), e.g., no more than 3 days total during the 2 week washout period, no more than 7 days total during the 4 week follow-up period. If a subject requires treatment for more than 7 days per month or requires systemic therapy, they may be discontinued from the study. Medications permitted are listed in Table 8.1.

In the event of an atopic dermatitis or pruritus exacerbation in between visits, subjects should contact study staff as soon as they are able. Subjects should seek approval on the use of rescue medications. In the event that the subject did not notify the study staff, every effort should be made by the subject to contact the PI or study staff as soon as feasible. The details of the medication should be recorded in the eDiary and transferred to the CRF. Details recorded should include medication name, date of administration, dosage, and number of applications.

**Table 8.1** Permitted Rescue Medication

| Class 4 – Mid-strength | |
|---|---|
| Clocortolone pivalate (0.1%) | Cloderm® Cream |
| Mometasone furoate (0.1%) | Elocon® Cream |
| Triamcinolone acetonide (0.1%) | Aristocort® A Cream, Kenalog® Ointment |
| Betamethasone valerate (0.1%) | Valisone Ointment |
| Fluocinolone acetonide (0.025%) | Synalar® Ointment |
| Class 5 – Lower Mid-strength | |
| Fluticasone propionate (0.05%) | Cutivate® Cream/Cutivate Lotion |
| Prednicarbate (0.1%) | Dermatop® Cream |
| Hydrocortisone probutate (0.1%) | Pandel® Cream |
| Triamcinolone acetonide (0.1%) | Aristocort A Cream, Kenalog Lotion |
| Fluocinolone acetonide (0.025%) | Synalar Cream |
| Class 6 – Mild | |
| Alclometasone dipropionate (0.05%) | Aclovate® Cream/Ointment |
| Desonide (0.05%) | Verdeso™ Foam, Desonate Gel™ |
| Triamcinolone acetonide (0.025%) | Aristocort A Cream, Kenalog Lotion |
| Hydrocortisone butyrate (0.1%) | Locoid Cream/Ointment |
| Fluocinolone acetonide (0.01%) | Derma-Smoothe/FS® Scalp Oil, Synalar Topical Solution |
| Class 7 – Least potent | |
| Hydrocortisone (2%/2.5%) | Nutracort® Lotion, Synacort Cream |
| Hydrocortisone (0.5 to 0.1%) | Cortaid® Cream/Spray/Ointment and many other over-the-counter products |

#### 8.14.2 Use of Excluded Therapies During the Treatment Period

Subjects who use an excluded therapy during the treatment period for treatment of atopic dermatitis or pruritus outside of the rescue medication allowance will be discontinued from study drug treatment, with the following exception:

• Subjects who require short treatment for indications other than atopic dermatitis or pruritus (up to a total of 3 days over the treatment period) with sedatives, tranquilizers, opioids, and/or topical therapies will not be required to discontinue from study drug treatment.

Use of any excluded therapies will be recorded for subjects who receive them.

#### 8.15 Handling of Investigational Product

Subjects will receive study IP in 30 ml white bottles. Each bottle will be anticipated for use over 10 days and brought to all study appointments. The IP bottle can be kept at room temperature while in use by the subject.

Subjects will be asked not to subject the treatment kit to conditions which are unnatural or harmful to the product, such as excessive heat (temperatures over 77°F (25°C)) and freezing temperatures (below 32°F (0°C)). Subjects may travel with their study medication but should not leave it in a hot car, outside in the cold temperatures, etc. Subjects will also be asked not to tamper or cause damage to IP.

#### 9 CONTRACEPTION REQUIREMENTS

Effective contraception is required for all women physiologically capable of becoming pregnant during study participation. Women of child-bearing potential must agree to use an acceptable form of contraception for up to 2 weeks after the study completion as detailed. Women of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile (e.g., by tubal ligation) or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.

Effective contraception methods include:

- Use of oral, injected or implanted hormonal methods of contraception or placement of an IUD or IUS or other forms of hormonal contraception that have comparable efficacy, for example hormone vaginal ring or transdermal hormone contraception
- Use of barrier methods (i.e., condom, diaphragm) used with a spermicide (i.e., foam, cream, or gel that kills sperm)
- Total abstinence (when this is in line with the preferred and usual lifestyle of the study participant).

Periodic abstinence (i.e., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.

Male participants of the study who are having sexual intercourse with a woman who can become pregnant must use an acceptable form of birth control while participating in the study. Additionally, male participants are expected to inform their female partners of their participation in a research study of an investigational drug, the effects of which on a fetus and on a pregnant woman are unknown. Male participants will also be expected to provide their female partners with the contraception requirements information previously described and the study doctor's contact information for questions.
Payment for all aspects of obstetrical care, child-or related care will be the study participant's responsibility.

In case of pregnancy, Investigational Product should be discontinued and the Sponsor should be informed immediately. Follow-up of the pregnancy will be mandatory until the outcome is available

#### 10 STUDY PROCEDURES

# **10.1 Pre-screening procedures**

Study subjects will be recruited from among participating hospitals, clinics, and diagnostic centers or from general population under the responsibility of a participating Investigator. Prior to initiation of the recruitment phase, participating Investigators will identify a pool of potential study subjects. Each of these centers will identify potentially eligible patients in advance, by either reviewing past medical records and diagnoses, screening in clinics, referral from other physicians, or other sources of recruitment, to identify those aged 18 to 65 with clinical diagnosis of mild or moderate Atopic Dermatitis. Medical records from patient's dermatologist or primary care physician to confirm the diagnosis are optional. Verbal confirmation of the diagnosis present for > 12 months is sufficient to fulfill this criterion.

#### 10.2 Informed Consent Procedures

Eligible participants may only be included in the study after providing a consent using the IRB-approved informed consent form. Informed consent must be obtained before conducting any study-specific procedures (i.e., all of the procedures described in the protocol). The process of obtaining informed consent should be documented in the participant's source documents. The date of signing of informed consent (and withdrawal, if later withdrawn) should be documented in the eCRF

#### **10.3 Study Assessments**

Study activities will take place according to the Time and Events table (Appendix A).

Demographics and a complete medical history will be recorded during the Screening period. The medical history will include a complete review of all current diseases and their respective durations and treatments

# 10.4 Inclusion procedures

Once all inclusion/exclusion criteria are fulfilled, the patient becomes eligible for randomization and inclusion into the treatment period. Treatment allocation will be performed as stated above

in Section 8.5. Study medication will be delivered as stated in Section 8.6. Patients will be counseled on product application and eDiary completion.

# 10.5 Timing of patient's visits to the clinic

Patients will be asked to report to the clinic for their scheduled appointments. If a subject is unable to schedule an appointment within the required time frame, study staff will be asked to reschedule the patient to a day when they are able to come in within predetermined time frame.

# 10.6 Description by type of visit

# **10.6.1** Screening Visit (-21 to -14) – Visit 1

- informed consent completed and signed
- inclusion and exclusion criteria
- demographic data
- medical/surgical history
- concomitant medications
- physical exam
- vital signs
- blood for clinical chemistry, serology and hematology
- urine pregnancy test (for women of childbearing potential)
- NRS assessment
- POEM questionnaire
- Pruritus 5-D questionnaire
- IGA scoring assessment
- EASI scoring assessment
- study counseling
- start eDiary
- start AE monitoring

# 10.6.2 Washout Phase (-14 to -1)

For those subjects who meet the eligibility criteria at the Screening visit and is determined by the Principal Investigator to be eligible for the study after the safety labs testing results are available, subjects will be notified by telephone to start the Washout period phase. Subjects will be allowed to use their regular emollients if needed but will be asked to stop using bleach or vinegar baths.

Stable doses of the following therapies for pruritus and/or atopic dermatitis will be allowed as adjunctive therapies during the study:

- Oral H1 antihistamines
- Bland emollients

A detailed guideline will be shared with the sites and subjects to ensure consistency in study medication treatment application and relation to body washing, emollient use, and other chemical exposure to skin.

Low- or mid-potency topical corticosteroids will be allowed per subjects' usual medication, frequency, and dose during the washout period but no more than 7 days per month as rescue medication.

Subjects using any of these adjunctive therapies should maintain their regimen without clinically significant changes in type, dose or frequency throughout the screening, treatment, and follow-up periods.

Subjects will be prohibited from using Excluded Medications/Therapy listed in Appendix B.

- phone call to subjects
- study counseling

# 10.6.3 Study Day 0-Baseline visit (0) – Visit 2

- inclusion and exclusion criteria
- concomitant medications
- medical history
- vital signs
- urine pregnancy test (for women of childbearing potential)
- NRS assessment
- POEM questionnaire
- Pruritus 5-D questionnaire
- IGA scoring assessment
- EASI scoring assessment
- allocation of a randomized treatment kit number via IWRS
- delivery of the corresponding Investigational Product
- obtain study medication weight for Investigational Product compliance
- first application of Investigational Product (under medical supervision)
- study counseling
- eDiary review
- recording of AEs if any

# 10.6.4 Day 5- Phone call to patient

The Day 5 visit is a telephone visit that occurs 5 days (±2 days) after the Baseline visit. Study staff will discuss IP application with the subject, answer any questions and counsel the subject on any other matters related to the study.

- phone call to subjects
- application of study drug
- study counseling

# 10.6.5 Day 14 and Day 28 study visits – Visit 3 and Visit 4

- concomitant medications
- vital signs
- blood for clinical chemistry and hematology (Day 28)
- urine pregnancy test (for women of childbearing potential) (Day 28)
- NRS assessment
- POEM questionnaire
- Pruritus 5-D questionnaire
- IGA scoring assessment
- EASI scoring assessment
- obtain study medication weight for Investigational Product compliance
- dispense investigational product to patient (Day 14)
- collect study medication
- application of study drug
- eDiary
- study counseling
- recording of AEs if any

# 10.6.6 Day 56-End of Study Visit – Visit 5

- concomitant medications
- vital signs
- physical exam
- urine pregnancy test (for women of childbearing potential)
- NRS assessment
- POEM questionnaire
- Pruritus 5-D questionnaire
- IGA scoring assessment
- EASI scoring assessment
- eDiary
- recording of AEs if any

# 10.6.7 Unscheduled/Unanticipated Study visit

If an event arises that requires patient to come in to the research center, subjects should be scheduled for the Unscheduled visit and assessments are performed based on investigator discretion.

# 10.6.8 Early Termination Visit

Every attempt should be made to complete all visits during the defined window periods. Subjects who do not complete all required study visits and withdraw from the study before the Day 56 final visit will be asked to complete the Early Termination Visit.

During the visit, the following will be obtained:

- concomitant medications
- vital signs
- physical exam
- urine pregnancy test (for women of childbearing potential)
- NRS assessment
- POEM questionnaire
- Pruritus 5-D questionnaire
- IGA scoring assessment
- EASI scoring assessment
- blood for clinical chemistry and hematology (if visit occurs before Day 28)
- eDiary
- collect study medication (if visit occurs before Day 28)
- obtain study medication weight for Investigational Product compliance
- recording of AEs if any

#### 11 STUDY ASSESSMENTS

#### 11.1 Safety Assessments

# 11.1.1 Vital Signs

Vital signs will include measurements of heart rate, sitting blood pressure, respiration rate, and temperature. Vital signs will be assessed as outlined in Appendix A and at unscheduled study visits when clinically indicated. The subjects' height and weight will be measured as outlined in Appendix A.

# 11.1.2 Physical Examinations

The physical examination will be performed at Screening, Day 56, and at any Unanticipated visit should one occur as outlined in Appendix A. The physical examination includes an assessment of general appearance and a review of systems (dermatologic, head, eyes, ears, nose, mouth/throat/neck, thyroid, lymph nodes, respiratory, cardiovascular, gastrointestinal, extremities, musculoskeletal, and neurologic systems).

### 11.1.3 Laboratory Assessments

Blood samples should be taken using standard venipuncture techniques. Blood sampling will be performed according to the site SOPs.

The following laboratory variables will be determined as outlined below:

The following routine clinical chemistry, hematology and Lipid Panel will be performed according to Time and Events table (Appendix A): Albumin, Alkaline Phosphatase, ALT, AST, Total Bilirubin, BUN, BUN: Creatinine ratio, Calcium, Chloride, Creatinine, eGFR, Glucose, Potassium, Sodium, Uric Acid, Total Protein, Bicarbonate

Lipid Panel: HDL Cholesterol, LDL cholesterol, Total Cholesterol, Triglycerides, VLDL Cholesterol, LDL/HDL Cholesterol Ratio, Non-HDL Cholesterol.

Urinalysis: Color, clarity, pH, specific gravity, bilirubin, glucose, ketones, leukocytes, nitrite, blood, protein, urobilinogen, microscopic analysis.

Hematology: WBC, RBC, Hemoglobin, Hematocrit, Platelets, WBC Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils)

Serology will only be done at Screening: HIV Ab, HCV Ab, and HBsAg.

Pregnancy testing: All females of childbearing potential will have a local urine pregnancy test performed at specified visits.

Patients will be asked to fast for at least 8 hours before all blood tests are done. An exception will be made on the laboratory testing for the screening visit such that either fasting or non-fasting blood samples can be collected. This is to avoid requesting participants to fast prior to the informed consent.

The total blood volume collected for clinical labs for Screening visit will be approximately 20 ml of whole blood. Volume collected for subsequent visits would be approximately 10 ml of whole blood.

Any value outside the normal range will be flagged for the attention of the Investigator or designee at the site. The Investigator or designee will indicate whether or not the value is of clinical significance. If the result of the clinical chemistry test from the samples taken during the screening phase is indicated as clinically significant, the study subject will NOT be allowed into the study.

### 11.2 Efficacy Assessments

Efficacy endpoints will be descriptively summarized and will include the number of observations, mean, median, standard deviation, minimum, and maximum of scores/values at all applicable time points and for all treatments in the ITT Population.

#### 11.2.1 EASI Assessment

An EASI score is used to measure the extent (area) and severity of atopic eczema (Eczema Area and Severity Index). The score will be calculated at the times indicated in the Time and Events Table (Appendix A). The investigator will assess improvement of eczema based on intensity and severity of the disease. EASI score sheet can be found in Appendix C.

The severity strata for the EASI are as follows:

0 = clear

0.1-1.0 = almost clear

 $1 \cdot 1 - 7 \cdot 0 = mild$ 

 $7 \cdot 1 - 21 \cdot 0 = moderate$ 

 $21 \cdot 1 - 50 \cdot 0 = \text{severe}$ 

 $50 \cdot 1 - 72 \cdot 0 = \text{very severe}$ 

#### 11.2.2 Patient Oriented Eczema Measure

The POEM is a tool developed by the University of Nottingham, United Kingdom, for monitoring atopic dermatitis severity (Appendix D). The subject will complete the questionnaire at each of the assessment timepoints as outlined in Appendix A.

Each of the 7 questions in the POEM questionnaire carries equal weight and is scored from 0 to 4:

- No days = 0.
- 1 to 2 days = 1.
- 3 to 4 days = 2.
- 5 to 6 days = 3.
- Every day = 4.

Scores are then added to yield a total score of 0 to 28; higher scores mean the greater the severity of atopic dermatitis.

# 11.2.3 Itch Numeric Rating Scale

The Itch NRS is a validated, self-reported instrument for measurement of itch intensity. It uses a 24-hour recall period and asks subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. In this study, both worst itch intensity (WI-NRS) and average itch intensity (AI-NRS) during a 24-hour recall period will be captured. Subjects will record their Itch NRS scores once

daily via eDiary throughout the screening, treatment, and follow-up periods, as outlined in Appendix A.

The question for WI-NRS would be, "Please rate the itching severity due to your atopic dermatitis by circling the number that best describes your worst level of itching in the past 24 hours."

The question for AI-NRS would be, "Please rate the itching severity due to your atopic dermatitis by circling the number that best describes your average level of itching in the past 24 hours."

0 1 2 3 4 5 6 7 8 9 10 0 = No itching 10 = Worst itch imaginable

# 11.2.4 Investigator Global Assessment Score (IGA)

IGA will be performed at the times indicated (Screening, Baseline, Day 14, Day 28, and Day 56) in the Time and Events Table of the Protocol (Appendix A) as static IGA. The Investigator will assess improvement of Atopic Dermatitis based on the 5-point severity scale summarized below and in Appendix E.

| Score | Category | Definition |
|---|---|---|
| 0 | Clear | Minor residual discoloration, no erythema or induration/papulation, no oozing/crusting |
| 1 | Almost Clear | Trace faint pink erythema with almost no induration/papulation and no oozing/crusting |
| 2 | Mild disease | Faint pink erythema with mild induration/papulation and no oozing/crusting |
| 3 | Moderate<br>disease | Pink-red erythema with moderate induration/papulation and there may be some oozing/crusting |
| 4 | Severe disease | Deep/bright red erythema with severe induration/papulation with oozing/crusting |

#### 11.2.5 5-D Pruritus Scale

The 5-D Pruritus Scale is a validated, multi-dimensional measure of itching that assesses the five domains of degree, duration, direction, disability and distribution (Appendix F). Subjects rate their symptoms over the preceding 2-week period on a 1 to 5 scale, with 5 being the most affected. Subjects will complete the 5-D Pruritus Scale during study visits as outlined in Appendix A.

# 11.3 eDiary and Efficacy Assessments

All patient reported outcomes and clinical outcome assessments (ePRO/eCOA) will be obtained electronically using either a smartphone application or a tablet. Participants will be provided with eDiary at screening to initiate daily diary entries from screening to follow-up and will include responses to WI-NRS, AI-NRS, daily dose confirmation (during the treatment period),

rescue medication (if any), and local skin tolerability (Day 1 to Day 7 of treatment). In addition, participants' usual adjunctive therapies (e.g., bland emollient, oral H-1 antihistamine) may be collected using eDiary or CRF at screening and optionally throughout the study. POEM and 5-D Pruritus Scale will be reported by the participants at the designated site visits using a site provided tablet. IGA and EASI will also be assessed at the designated site visits by the clinician.

# 11.4 Patient Reported Local Tolerability

Solicited local adverse reactions (e.g., itching, new rash, pain, tenderness, stinging, skin color change, etc.) and severity from subjects will be collected during the first week of treatment using eDiary with the questions outlined in Appendix G to inform local skin tolerability.

### 11.5 Pregnancy Reporting

Any pregnancy will be reported by study participants during their study participation. Participants who report pregnancy or lactation during the review of inclusion/exclusion criteria prior to randomization will not be enrolled in the trial. In case of pregnancy, Investigational Product should be discontinued and the Sponsor informed. Follow-up of the pregnancy will be mandatory until the outcome is available.

# 11.6 Study Completion

A completed participant is one who has completed all study visits. Day 56 study visit is defined as the participant's last visit.

# 11.7 Subject Withdrawal Criteria

A subject may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the Investigator for safety, behavioral, or administrative reasons.

Reasons for withdrawal (subjects who refuse to return for any remaining study visits) or discontinuation (subjects who prematurely stop the application) at any time during the study may include, but are not limited, to the following:

- For safety reasons, either at the discretion of the Investigator or at the subject's request
- For protocol violations at the discretion of AOBiome
- Due to concomitant therapy that could interfere with the results of the study (the Investigator will report all such information on the CRFs and decide, in accordance with AOBiome, whether the subject is to be withdrawn).

All premature discontinuations and their causes must be carefully documented by the Investigator on the CRF or if needed on the AE form.

If, for any reason, a subject is withdrawn before completing the final visit, the reason for termination will be entered on the CRF. All data gathered on the subject prior to termination will

be made available to AOBiome. Subjects not completing the entire study should be fully evaluated when possible. The appropriate CRFs should be completed.

If the subject chooses to withdraw before completing the study, the subject should notify the study coordinator who will instruct the subject on completion of assessments for End of Study (EOS) visit. For subjects who refuse to complete the assessments for their early termination, every attempt must be made to check on their status, using any mode of communication such as telephone, email, fax, or text.

# 12 STATISTICAL CONSIDERATIONS

# 12.1 Sample Size

Approximately 576 subjects may be enrolled to account for 16.7% drop out rate prior to completing the study. A total of 160 evaluable subjects per group (480 total) are required to achieve at least 80% power to detect a pairwise difference of 0.65 in mean WI-NRS change from baseline to Week 4 between one of two active doses of B244 and vehicle control when assuming a standard deviation of 2.5 and applying a Dunnett Testing Method at a one-sided familywise error rate of 0.10.

### 12.2 Populations for Analysis

Intent to Treat (ITT): All randomized participants who apply at least 1 dose of study medication. Subjects will be grouped as randomized.

Per Protocol: All subjects in the ITT population without any major protocol deviations that may have an impact on the efficacy assessments, who complete their Week 4 visit, and who administer at least 50% of investigational product (IP). Subjects will be grouped as treated.

Safety: All subjects who apply at least 1 dose of study medication. Subjects will be grouped as treated.

# 12.3 Data Analysis

A separate statistical analysis plan will be developed. All data collected will be documented using summary tables, figures, and/or patient data listings. For continuous variables, descriptive statistics (number (n), mean, median, standard deviation, minimum and maximum) will be presented. For categorical variables, frequencies and percentages will be presented. As appropriate, a 95% CI will be presented. Graphical displays will be presented, as appropriate. Data will be presented by treatment group and overall.

Descriptive statistics for each treatment group will be provided for clinical laboratory values (e.g., hematology, serum chemistry, and urinalysis) and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation. Abnormal clinical laboratory values will be listed.

### 12.3.1 Disposition

A tabulation of the disposition of subjects will be presented, including the number enrolled, the number randomized, the number treated, and the reasons for study discontinuation. Summaries of the number in each analysis set will be presented. Entry criteria violations and protocol deviations will be listed.

# 12.3.2 Demographic and Baseline

Demographic and baseline characteristic data summarization will be performed in order to descriptively assess the comparability of treatment groups. Data to be tabulated will include age, race, ethnicity, height, weight, and BMI, as well as baseline characteristics related to medical history.

### 12.4 Safety Analyses

#### 12.4.1 Definitions

All adverse events recorded during the study will be coded according to MedDRA.

#### 12.4.2 Adverse Events

All adverse events (AEs) recorded during the study through the date of randomization through 28 days after the last dose of study drug will be analyzed.

Adverse events will be summarized by treatment group using the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment-emergent AEs (TEAEs), treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, discontinuations due to AEs, and AEs  $\geq$  Grade 3 severity. By-subject listings will be provided for any deaths, SAEs, and AEs leading to discontinuation.

AE's will be summarized using incidence rates. Therefore, each subject will only contribute once for a given adverse event SOC or PT.

Any treatment emergent AEs related to local safety (e.g., erythema, edema, induration, vesiculation, etc.) will be collected by the investigator during scheduled clinic visits. In addition, solicited local adverse reactions (e.g., itching, new rash, pain, tenderness, stinging, skin color change, etc.) and severity from subjects will be collected during the first week of treatment using eDiary to inform local skin tolerability.

A summary of the incidence of any adverse event, SAE, and adverse events leading to discontinuation will be presented. Summaries will display, by treatment group, the incidence of patients with events, the frequency of patients with events within each primary system organ class and by preferred terms. For each preferred term and each system organ class a patient will

be counted only once. For summaries on severe or drug-related AE, for a given patient, the highest severity or relationship for a specific preferred term will be considered.

#### 12.4.3 Deaths and Serious Adverse Events

Serious adverse events and events leading to death will be summarized overall and by primary system organ class and preferred term.

# 12.4.4 Adverse Events leading to treatment discontinuation

Adverse events leading to treatment discontinuation will be summarized overall and by primary system organ class and preferred term.

# 12.5 Efficacy Analyses

All efficacy analyses will be performed on the ITT population and PP population. Regression models will include all eligible subjects for the respective analysis, from the 3 treatment arms.

Hypothesis tests for the primary efficacy endpoint will be performed using a Dunnett Testing Method, applying pairwise comparisons of each respective B244 dose group to vehicle using a one-sided familywise error rate of 0.10. No additional adjustments will be made for multiple testing. As such, p-values from analysis of secondary and exploratory efficacy analyses must be interpreted in an exploratory fashion.

The primary endpoint of mean change from baseline to Week 4 in WI-NRS will be analyzed using analysis of covariance (ANCOVA) models.

In addition, continuous efficacy endpoints will be summarized using descriptive statistics at Baseline, Week 2, Week 4 and Week 8 for actual values and change-from-baseline values. The difference in treatment groups in change-from-baseline values at post-baseline visits will be analyzed using a mixed model with repeated measures to account for within subject variability and including visit (Baseline vs. Week 2, Week 4, Week 8), treatment group, visit-by-treatment interaction, and baseline value as explanatory variables.

Categorical variables will be summarized using descriptive statistics and analyzed using a logistic regression model at each respective timepoints. Generalized estimating equations to account for repeated measures and within-subject variability may also be applied.

Supportive analyses may be performed combining the B244 dose groups in comparison against vehicle and comparison of the B244 groups to one another.

### 12.6 Handling of dropouts or missing data

All available data will be analyzed. The details for any imputations for missing data will be documented in the trial's Statistical Analysis Plan. Subjects who dropout after enrollment but prior to randomization will be replaced.

#### 12.7 Clinical Trial Protocol deviations

At minimum, the following deviations will be summarized on the ITT patient population:

- Inclusion or exclusion criteria not satisfied.
- Deviations related to the Investigational Product administration
- Not permitted concomitant medications.

# 13 ADVERSE EVENTS (AE) AND SERIOUS ADVERSE EVENTS (SAE)

The Investigator and study staff are responsible for detecting and recording AEs and SAEs during scheduled safety evaluations and whenever such information is brought to their attention. This section of the protocol provides definitions and detailed procedures to be followed.

#### 13.1 Definition of an AE

An AE is any untoward medical occurrence in a study participant which is temporally associated with the use of a medicinal product, regardless of its potential relationship to the medicinal product. An AE, therefore, can be any unfavorable or unintended sign, including an abnormal symptom, or disease (new or exacerbated), whether or not related to the investigational product (IP).

Examples of an AE include:

- Exacerbation of a pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after investigational product administration even though it may have been present prior to the start of the study.
- Signs, symptoms of a drug interaction.
- Signs, symptoms of a suspected overdose of either investigational product or a concurrent medication (overdose per se should not be reported as an AE/SAE).

AEs may include pre- or post-treatment events that occur as a result of protocol-mandated procedures (i.e., modification of participant's previous therapeutic regimen).

### 13.2 Definition of a SAE

A serious adverse event is any untoward medical occurrence that, at any dose:

- a) results in death.
- b) is life-threatening.

NOTE: The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

c) requires hospitalization or prolongation of existing hospitalization.

NOTE: In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or out -patient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious. Routine hospitalizations or elective surgeries are generally not regarded as SAEs.

d) results in disability/incapacity

NOTE: The term disability means a substantial disruption of a person's ability to conduct normal life functions. This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g. sprained ankle) which may interfere or prevent everyday life functions but do not constitute a substantial disruption.

- e) is a congenital anomaly/birth defect
- f) Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These should also be considered serious. Examples of such events are invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

# 13.3 Time-period, Frequency, and Method of Detecting AEs and SAEs

All AEs occurring after administration of the first dose of study medication and on or before the final assessment must be reported as AEs. All AEs must be recorded irrespective of whether they are considered drug-related.

At each assessment in the period defined above, AEs will be evaluated by the Investigator and recorded.

Any AEs already documented at a previous assessment and designated as ongoing, should be reviewed at subsequent assessments as necessary. If these have resolved, this should be documented. Changes in intensity or frequency of AEs should be recorded as separate events (i.e., a new record started).

The recording of AEs and SAEs are described in Section 13.4 ("Recording of AEs and SAEs").

# 13.4 Recording of AEs and SAEs

All clinical events, including either observed or volunteered problems, complaints or symptoms are to be recorded on the Adverse Events page(s) of the CRF. The need to capture this information is not dependent upon whether the clinical event is associated with study treatment. Adverse clinical events resulting from concurrent illnesses or reactions to concurrent medications are also to be recorded. In order to avoid vague, ambiguous, or colloquial expressions, the AE should be recorded in standard medical terminology rather than the participant's own words.

Each adverse clinical event is to be evaluated for duration, intensity, and whether the event may be associated with the investigational product (IP) or other causes. Start and stop dates, relationship to investigational product (IP), medical management, and alternative causality of event must be recorded in the Adverse Events section of the CRF. AEs believed to be possibly related to investigational product (IP) must be followed until resolution.

# 13.5 Evaluating AEs and SAEs

# 13.5.1 Severity Rating

The severity of an adverse event (AE and SAE) is to be scored according to the following scale:

| Mild | Awareness of symptoms, but easily tolerated |
|----------|-----------------------------------------------------------------|
| Moderate | Discomfort enough to cause interference with usual activity |
| Severe | Incapacitating with inability to work or perform usual activity |

An AE that is assessed as severe should not be confused with a SAE. An event is defined as 'serious' when it meets one of the pre-defined outcomes as described in Section 13.2 "Definition of a SAE".

### 13.5.2 Relationship to Investigational product (IP)

SAEs will be classified as "not related" or "related" (including unknown).

<u>For AEs</u>, the relationship to study treatment is to be assessed according to the following definitions:

**Definitely not related:** The AE is definitely not related to the drug. This designation should be reserved for those events which occur prior to study treatment or for those events which cannot be even remotely related to study participation (e.g., injuries sustained in an automobile accident).

**Unlikely related:** There is no reasonable association between the study treatment and the suspected event and the event could have been produced by the participant 's clinical state or other modes of therapy administered to the participant.

**Possibly related:** The suspected adverse event may or may not follow a reasonable temporal sequence from study treatment administration but seems to be the type of reaction that cannot be dismissed as unlikely. The event could have been produced or mimicked by the participant 's clinical state or by other modes of therapy concomitantly administered to the participant.

**Probably related:** The suspected adverse event follows a reasonable temporal sequence from study treatment administration, abates upon discontinuation of the treatment, and cannot be reasonably explained by the known characteristics of the participant 's clinical state.

**Definitely related**: This designation should be reserved for those events which have no uncertainty in their relationship to treatment administration.

#### 13.6 Pregnancy

Any pregnancy that occurs in a female participating in the study must be reported to the Safety Team or to a designated Safety email or fax number provided by the Safety Team within 24 hours of learning of the pregnancy. Follow-up must occur to determine the outcome of the pregnancy (including premature termination) and the status of mother and child. Pregnancy complications and elective terminations for medical reasons must be reported as AEs or SAEs. Spontaneous abortions must be reported as an SAE.

Any SAE occurring in association with a pregnancy and considered by the Investigator as related to the investigational product must be promptly reported to the Sponsor, even if the event occurred after the participant completed the study.

The Investigator must attempt to collect pregnancy information on any female partners of male participants who become pregnant while the male participant is enrolled in the study. Pregnancy information must be reported to the Sponsor as described above.

#### 13.7 Prompt Reporting of SAEs to the Sponsor

In the case of a Serious Adverse Event the Investigator must immediately:

- **SEND** (within 1 working day) the signed and dated SAE Report Form to the Safety Team or to a designated Safety email or fax number provided by the Safety Team;
- ATTACH a photocopy of all examinations carried out and the dates on which these
  examinations were performed. Care should be taken to ensure that the patient's identity is
  protected and the patient's identifiers in the Clinical Trial are properly documented on all
  copies of source documents provided to the Sponsor. For laboratory results, include the
  laboratory normal ranges;
- Follow-up of any Serious Adverse Event that is fatal or life threatening should be provided within one additional calendar week. The treatment code will be unblinded for reporting of Serious Adverse Events that are unexpected and determined to be related to the use of the Investigational Product.

# Follow-up

- The Investigator should take all appropriate measures to ensure the safety of the patients, including referral to a specialist if indicated. Notably the Investigator should follow up the outcome of any adverse events (clinical signs, laboratory values or other, etc.) until the return to normal or stabilization of the patient's condition;
- In the case of any Serious Adverse Event, the patient must be followed up until clinical recovery is complete and laboratory results have returned to normal, or until progression has been stabilized. This implies that follow-up may continue after the patient has left the Clinical Trial and that additional investigations may be requested by the Safety Team;
- In case of any Serious Adverse Event brought to the attention of the Investigator at any time after cessation of Investigational Product and considered by the Investigator to be related to the Investigational Product, this should be reported to the Safety Team.

# **AOBiome Reportable Events Hotline**

Email: safety@aobiome.com

#### 14 ETHICAL AND REGULATORY STANDARDS

#### 14.1 Ethical Conduct of Study

This clinical trial was designed and shall be implemented, executed, and reported in accordance with the ICH Harmonized Tripartite Guidelines for Good Clinical Practice, with applicable local

regulations (including US Code of Federal Regulations Title 21), and with the ethical principles laid down in the Declaration of Helsinki.

The Investigator(s) should conduct the study in accordance with this protocol, the Declaration of Helsinki and ICH GCP guidelines and FDA regulations. The Investigator(s) and the Sponsor will sign the protocol and study contract, to confirm agreement. The Investigator(s) will not implement any amendment (deviation or changes of the protocol) without agreement by the Sponsor and IRB approval, except where necessary to eliminate immediate hazard(s) to study participants, or when change(s) involve only logistical or administrative aspects of the study. Records that may reveal the identities of participants must be well protected, with consideration given to confidentiality and the right to privacy of participants.

# 14.2 Laws and Regulations

This Clinical Trial will be conducted in compliance with all international laws and regulations, and national laws and regulations of the countries in which the clinical trial is performed, as well as any applicable guidelines. The trial will be registered and updated on www.clintrials.gov and on other sites, as deemed appropriate.

#### 14.3 Informed Consent

Each participant must be provided with a statement that the investigation involves research and that the IRB has approved solicitation of participants to participate; a fair explanation of the procedures to be followed and their purposes, including identification of any procedures which are experimental; a description in lay language of any possible side effects; a description of any attendant discomforts and risks reasonably to be expected; a description of any benefits reasonably to be expected; a disclosure of any appropriate alternative procedures that might be advantageous for the participant; an offer to answer any inquiries concerning the procedures, and instruction that the person is free to withdraw consent and discontinue participation in the project or activity at any time without prejudice to the participant. Payment to research participants for taking part in the study is based on time and inconvenience. All information concerning payment, including the schedule of payments, must be set forth in the informed consent, including a disclosure that the Investigator is being paid to perform the stated research.

A participant must give consent to take part in the study. Participants below the age of majority in the municipality must give written assent to participate in this study. This consent must be dated and retained by the Principal Investigator as part of the study records. A downloadable digital copy shall be given to the person signing the form. The informed consent process must be documented in the participant's source documents.

The Investigator agrees that the Sponsor, its employees or agents will have the right from time to time during the course of this study to audit and review pertinent medical records relating to this clinical trial. A statement will be obtained from each person participating in the study permitting the release of his/her medical records as necessary for inspection by authorized personnel of the Sponsor, FDA, and the staff managing the clinical study.

The release of medical records and the review of the contents will be in compliance with the Health Insurance Portability and Accountability Act of 1996 (HIPAA).

# 14.4 Institutional Review Board/Independent Ethics Committee (IRB/EC)

The protocol and informed consent form and the electronic version of the consent for this study must be approved by the IRB. A copy of the Letter of Approval from the Board, which contains specific identification of the documents approved, must be received by the Sponsor prior to shipment of drug supplies to the Principal Investigator.

All changes to the protocol, as well as a change of Investigator, must also be approved by the IRB and documentation of this approval provided to the study monitor. Records of the IRB's review and approval of all documents pertaining to the study must be kept on file by the Principal Investigator and are subject to FDA inspection at any time. IRB renewal for approval is required each year. The Investigator is to inform AOBiome, in writing, of the approval to continue the study.

# 14.5 Clinical Monitoring/Record Keeping

There shall be no alterations in the protocol design without the written consent and approval of the Sponsor and the approval of the IRB, except in the case that participants are at immediate risk without immediate implementation of such alterations. In the aforementioned situation, the site should notify the Sponsor and IRB of the deviation as soon as possible, and should seek the written consent and approval of the Sponsor and the approval of the IRB.

All results of this trial must be recorded on eCRFs. Each participant who has been randomized must have a completed eCRF. Reasons for termination must be stated in the early termination section. Study participants are not to be identified by name on eCRFs, but rather by coded identifiers and participant initials.

The study monitor will verify the accuracy of the data by reviewing pertinent source documents such as office records or hospital charts of the participants.

Study records include eCRFs, signed FDA Form 1572, original reports of test results, and signed electronic informed consent forms. IRB approval letters and other documents pertaining to the conduct of the study are to be kept on file by the Investigator. If the study files are assigned to someone else or removed to another location, the Investigator is to notify the study monitor or Sponsor in writing of the change. All study records are subject to FDA inspection at any time. All information supplied to the Investigator by the Sponsor before, during, and after the study is confidential. Such information is to be used solely in connection with the clinical study. The study protocol, IB, and any other pertinent study related materials or records provided are to be maintained in a confidential manner, reviewed carefully with attention to admonitions and

returned to the Sponsor upon request. No part of these materials may be reproduced or transmitted in any form without prior written permission from the Sponsor.

#### 15 ADMINISTRATIVE RULES

#### 15.1 Curriculum Vitae

An updated, signed, and dated copy of the curriculum vitae with the experience, qualifications and training for each Investigator and/or Sub-Investigator(s) will be provided to the Sponsor prior to the beginning of the Clinical Trial.

# 15.2 Archiving of Study Documentation

The Investigator must maintain confidentiality for all study documentation, and take measures to prevent accidental or premature destruction of these documents.

It is recommended that the Investigator retain the study documents at least fifteen (15) years after the completion or discontinuation of the Clinical Trial. However, applicable regulatory requirements should be taken into account in the event that a longer period is required.

The Investigator must notify the Sponsor prior to destroying any study essential documents within the fifteen (15) year period following the Clinical Trial completion or discontinuation. If the Investigator's personal situation is such that archiving can no longer be ensured by him/her, the Investigator shall inform the Sponsor and the relevant records shall be transferred to a mutually agreed upon designee.

### 15.3 Internal Safety Review Committee

An internal safety review committee may be set up as needed to protect the ethical and safety interests of participants and to protect the scientific validity of the study. Ad-hoc safety interim analyses might be performed by an independent statistician if the safety review committee identifies potential safety signals during its routine blinded safety review. The details for the analysis plan may be documented in the trial's Statistical Analysis Plan.

#### 16 STUDY MONITORING

# **16.1** Responsibilities of the Investigator(s)

The Investigator(s) undertake(s) to perform the Clinical Trial in accordance with this Clinical Trial Protocol, ICH guidelines for Good Clinical Practice and the applicable regulatory requirements.

The Investigator is required to ensure compliance with all procedures required by the Clinical Trial Protocol and by study procedures provided by the Sponsor (including security rules). The Investigator agrees to provide reliable data and all information requested by the Clinical Trial Protocol (with the help of the Case Report Form [CRF], Discrepancy Resolution Form [DRF] or

other appropriate instrument) in an accurate and legible manner according to the instructions provided and to ensure direct access to source documents to Sponsor representatives. If any particular circuits have to be defined (e.g., e-CRF, Fax), particular attention should be paid to the confidentiality of the patient's data to be transferred. The Investigator may appoint such other individuals as he/she may deem appropriate as Sub-Investigators to assist in the conduct of the Clinical Trial in accordance with the Clinical Trial Protocol. All Sub-Investigators shall be timely appointed and listed. The Sub-Investigators will be supervised by and under the responsibility of the Investigator. The Investigator will provide them with a Clinical Trial Protocol and all necessary information.

### 16.2 Responsibilities of the Sponsor

The Sponsor of this Clinical Trial is responsible to Health Authorities for taking all reasonable steps to ensure the proper conduct of the Clinical Trial Protocol with regard to ethics, Clinical Trial Protocol compliance, integrity and validity of the data recorded on the Case Report Forms. Thus, the main duty of the Monitoring Team is to help the Investigator and the Sponsor maintain a high level of ethical, scientific, technical and regulatory quality in all aspects of the Clinical Trial. At regular intervals during the Clinical Trial, the site will be contacted, through monitoring visits, letters or telephone calls, by a representative of the Monitoring Team to review study progress, Investigator and patient compliance with Clinical Trial Protocol requirements, and any emergent problems. During these monitoring visits, the following but not exhaustive list of points will be scrutinized with the Investigator: patient informed consent, patient recruitment and follow-up, Serious Adverse Event documentation and reporting, outcome events documentation and reporting, Investigational Product allocation, patient compliance with the Investigational Product regimen, Investigational Product accountability, concomitant therapy use and quality of data.

#### 16.3 Source document requirements

According to the ICH guidelines for Good Clinical Practice, the Monitoring Team must check the Case Report Form entries against the source documents. The Informed Consent Form will include a statement by which the patient allows the Sponsor's duly authorized personnel, the Ethics Committee (IRB/EC), and the regulatory authorities to have direct access to source data which supports the data on the Case Report Forms (e.g., patient's medical file, appointment books, original laboratory records, etc.). These personnel, bound by professional secrecy, must keep confidential all personal identity or personal medical information (according to confidentiality rules).

#### 16.4 Use and completion of Case Report Forms (CRFs) and additional requests

The sponsor or CRO will be responsible for activities associated with the data management of this study. This will include setting up a relevant database and data transfer mechanisms, along with appropriate validation of data and resolution of queries. Data generated within this

clinical study will be handled according to the relevant SOPs of the data management and biostatistics departments of sponsor or CRO.

For Electronic Data Capture (EDC):

Study sites will enter data directly into an EDC system by completing the eCRF via a secure internet connection. Data entered into the eCRF must be verifiable against source documents at the study site. Any changes to the data entered into the EDC system will be recorded in an automated, secure audit trail and is Food and Drug Administration (FDA) Code of Federal Regulations (CFR) Title 21 Part 11 compliant.

Data entered into the eCRF will be validated as defined in the Data Validation Specifications (DVS). Validation includes, but is not limited to, validity checks (for example, missing data, range checks) and consistency checks (logical checks between variables) to ensure that study data are accurately reported. Additionally, CRO Data Management will perform aggregate data review as defined in the DVS to ensure that the data are complete, consistent and reasonable. The electronic edit checks will run continually throughout the course of the study and queries reviewed by CRO personnel to assure validity as compared to source records. Manual queries may also be entered into EDC by Monitoring or Data Management personnel to address identified discrepancies.

Medical conditions/procedures will be coded using MedDRA and prior and concomitant medications will be coded using WHODrug.

At the conclusion of the study, each site will be provided with their subject CRFs in Portable Document Format (PDF) for archival. The CRF PDFs will contain subject data, audit trail information, queries including responses, and comments.

### 17 PUBLICATIONS

All data generated from this study are the property of AOBiome LLC and shall be held in strict confidence along with all information furnished by AOBiome. Independent analyses and/or publication of these data by the Investigator or any member of his/her staff is not permitted without prior written consent of AOBiome.

Any formal presentation or publication of data from this trial will be considered as a joint publication by the Investigator(s) and appropriate Sponsor personnel. Authorship will be determined by mutual agreement. Written permission to the Investigator will be contingent on the review by the Sponsor of the methodology and statistical analysis and any publication or presentation will provide for nondisclosure of AOBiome confidential or proprietary information. In all cases, the parties agree to submit all manuscripts or abstracts to all other parties at least 30 days prior to submission. This will enable all parties to protect proprietary information and to provide comments based on information that may not yet be available to other parties.

#### 18 PROTOCOL ADHERENCE

This protocol defines the study objectives, the study procedures and the data to be collected on study participants. Additional assessments required to ensure the safety of participants should be administered as deemed necessary on a case by case basis. Under no circumstances is an Investigator allowed to collect additional data or conduct any additional procedures for any research related purpose involving any investigational drugs under the protocol. Investigators ascertain they will apply due diligence to avoid protocol deviations. If an Investigator feels a protocol deviation would improve the conduct of the study this must be considered a protocol amendment, and unless such an amendment is agreed upon by the sponsor and approved by the IRB/IEC and health authorities, where required, it cannot be implemented.

#### 19 CLINICAL TRIAL PROTOCOL AMENDMENTS

Any protocol amendments will be added as stand-alone documents. In addition, any and all revisions dictated by the amendments will be made in the protocol. Each time a protocol is amended, a new amended version date will be added to the cover page.

The Investigator should not implement any deviation from, or changes of the Clinical Trial Protocol without agreement by the sponsor and prior review and documented approval/favorable opinion from the IRB/EC of an amendment. The Investigator is expected to take any immediate action required for the safety of any participant included in this study, even if this action represents a deviation from the protocol. In such cases, the reporting requirements identified in Section 13 must be followed and the Study Lead.

#### 20 CONFIDENTIALITY

All information disclosed or provided by the Sponsor (or any company/institution acting on their behalf), or produced during the Clinical Trial, including, but not limited to, the Clinical Trial Protocol, the CRFs, the Investigator's Brochure and the results obtained during the course of the Clinical Trial, is confidential. The Investigator or any person under his/her authority agrees to undertake to keep confidential and not to disclose the information to any third party without the prior written approval of the Sponsor. However, the submission of this Clinical Trial Protocol and other necessary documentation to the Ethics Committee (IRB/EC) is expressly permitted, the IRB/EC members having the same obligation of confidentiality. The Sub-Investigators shall be bound by the same obligation as the Investigator. The Investigator shall inform the Sub-Investigators of the confidential nature of the Clinical Trial. The Investigator and the Sub-Investigators shall use the information solely for the purposes of the Clinical Trial, to the exclusion of any use for their own or for a third party's account.

#### 21 PROPERTY RIGHTS

All information, documents and Investigational Product provided by the Sponsor or its designee are and remain the sole property of the Sponsor. The Investigator shall not mention any information or the Product in any application for a patent or for any other intellectual property rights. All the results, data, documents and inventions, which arise directly or indirectly from the

Clinical Trial in any form, shall be the immediate and exclusive property of the Sponsor. The complete verified database will be shared with the Operations Committee, which shall have full access to all data. The Sponsor may use or exploit all the results at its own discretion, without any limitation to its property right (territory, field, continuance). The Sponsor shall be under no obligation to patent, develop, market or otherwise use the results of the Clinical Trial. As the case may be, the Investigator and/or the Sub-Investigators shall provide all assistance required by the Sponsor, at the Sponsor's expense, for obtaining and defending any patent, including signature of legal documents.

# 22 DATA PROTECTION

The patient's personal data and Investigator's personal data which may be included in the Sponsor database shall be treated in compliance with all applicable laws and regulations;

When archiving or processing personal data pertaining to the Investigator and/or to the patients, the Sponsor shall take all appropriate measures to safeguard and prevent access to this data by any unauthorized third party.

#### 23 SPONSOR AUDITS AND INSPECTIONS BY REGULATORY AGENCIES

For the purpose of ensuring compliance with the Clinical Trial Protocol, Good Clinical Practice and applicable regulatory requirements, the Investigator should permit auditing by or on behalf of the Sponsor and inspection by applicable regulatory authorities.

The Investigator agrees to allow the auditors/inspectors to have direct access to his/her study records for review, being understood that these personnel are bound by professional secrecy, and as such will not disclose any personal identity or personal medical information.

The Investigator will make every effort to help with the performance of the audits and inspections, giving access to all necessary facilities, data, and documents. As soon as the Investigator is notified of a future inspection by the authorities, he will inform the Sponsor and authorize the Sponsor to participate in this inspection.

The confidentiality of the data verified and the protection of the patients should be respected during these inspections.

Any result and information arising from the inspections by the regulatory authorities will be immediately communicated by the Investigator to the Sponsor.

The Investigator shall take appropriate measures required by the Sponsor to take corrective actions for all problems found during the audit or inspections.

# 24 PREMATURE DISCONTINUATION OF THE STUDY OR PREMATURE CLOSE-OUT OF A SITE

# 24.1 Decided by the Sponsor in the following cases:

- 1. In the event the results of the Clinical Trial do not appear to be scientifically convincing to the Sponsor;
- 2. If the aim of the Clinical Trial has become outdated or is no longer of interest;
- 3. If the information on the product leads to doubt as to the benefit/risk ratio;
- 4. If the Investigator has received from the Sponsor all Investigational Product, means and information necessary to perform the Clinical Trial and has not included any patient after a reasonable period of time mutually agreed upon;
- 5. In the event of breach by the Investigator of a fundamental obligation under this agreement, including but not limited to breach of the Clinical Trial Protocol, breach of the applicable laws and regulations or breach of the ICH guidelines for GCP;
- 6. If the total number of patients are included earlier than expected; In any case the Sponsor will notify the Investigator of its decision by written notice.

# 24.2 Decided by the Investigator

The Investigator must notify (30 days' prior notice) the Sponsor of his/her decision and give the reason in writing. In all cases (decided by the sponsor or by the Investigator), the appropriate Ethics Committee(s) (IRB/EC) and Health Authorities should be informed.

# 25 CLINICAL TRIAL PROTOCOL AMENDMENTS

All appendices attached hereto and referred to herein are made part of this Clinical Trial Protocol. The Investigator should not implement any deviation from, or changes of the Clinical Trial Protocol without agreement by the sponsor and prior review and documented approval/favorable opinion from the IRB/EC of an amendment, except where necessary to eliminate an immediate hazard(s) to clinical trial patients, or when the change(s) involves only logistical or administrative aspects of the trial. Any change agreed upon will be recorded in writing, the written amendment will be signed by the Investigator and by the Sponsor and the signed amendment will be filed with this Clinical Trial Protocol. Any amendment to the Clinical Trial Protocol requires written approval/favorable opinion by the IRB/EC prior to its implementation, unless there are overriding safety reasons. In some instances, an amendment may require a change to the Informed Consent Form. The Investigator must receive an IRB/EC approval/favorable opinion concerning the revised Informed Consent Form prior to implementation of the change.

#### **26 REFERENCES**

- 1. Eichenfield LF, Tom WL, Chamlin SL, et al. Guidelines of care for the management of atopic dermatitis: Section 1: Diagnosis and assessment of atopic dermatitis. *J Am Acad Dermatol*. 2014; 70(2):338-351.
- 2. Arp DJ, Sayavedra-Soto LA, Hommes NG. Molecular biology and biochemistry of ammonia oxidation by Nitrosomonas europaea. *Arch Microbiol* 2002; 178: 250-255.
- 3. Chandran K, Stein LY, Klotz MG, van Loosdrecht MCM. Nitrous oxide production by lithotrophic ammonia-oxidizing bacteria and implications for engineered nitrogen-removal systems. *Biochem Soc Trans* 2011; 39: 1832-1837.
- 4. Williams HC, Dellavalle RP, Garner S. Acne vulgaris. *The Lancet* 2012; 379(9813): 361-372. doi:10.1016/S0140-6736(11)60321-8.
- 5. Weller R, Price RJ, Ormerod AD, Benjamin N, & Leifert C. Antimicrobial effect of acidified nitrite on dermatophyte fungi, Candida and bacterial skin pathogens. *Journal of Applied Microbiology* 2001; *90*(4): 648-652.
- 6. Rico J, Quiring J, Hollenbach S, Enloe C, & Stasko N. Phase 2 study of efficacy and safety of SB204 in the treatment of acne vulgaris. *J Invest Dermatology* 2014; 134(8): S8.
- 7. Williams H, Robertson C, Stewart A, et al. Worldwide variations in the prevalence of symptoms of atopic eczema in the international study of asthma and allergies in childhood. *J Allergy Clin Immunol* 1999; 103: 125–138.
- 8. Diepgen, TL. Is the prevalence of atopic dermatitis increasing? In: Williams HC ed. Atopic Dermatitis: the Epidemiology, Causes and Prevention of Atopic Eczema. 2000 Cambridge: Cambridge University Press.
- 9. Roekevisch E, Spuls PI, Kuester D, Limpens J, Schmitt J. Efficacy and safety of systemic treatments for moderate-to-severe atopic dermatitis: a systematic review. *J Allergy Clin Immunol* 2014; 133(2):429-38.
- 10. Kobayashi T, Glatz M, Horiuchi K, Kawasaki H, Akiyama H, Kaplan DH, Kong HH, Amagai M, Nagao K. Dysbiosis and Staphylococcus aureus Colonization Drives Inflammation in Atopic Dermatitis. *Immunity* 2015; 42(4):756-66.

# **APPENDIX A: SCHEDULE OF EVENTS**

| Visit Name | Screening | Washout phase | Baseline Day 0 | Day 5 | Day 14<br>(Week 2) | Day 28<br>(Week 4) | Day 56<br>(Week 8) | Early<br>Termination<br>Visit | Comments/Clarification |
|---|---|---|---|---|---|---|---|---|---|
| Visit Number | V1 | | V2 | | V3 | V4 | V5 | | |
| Visit Window in days | -21 to -14 | -14 to -1 | 0 | +/-2 | +/-2 | +/-2 | +/-3 | | |
| Informed<br>Consent | X | | | | | | | | Informed consent will occur prior to any protocolmandated procedures, including the stopping of any excluded therapies. |
| Inclusion / Exclusion Criteria | X | | X | | | | | | |
| Demographics | X | | | | | | | | |
| Medical History | X | | X | | | | | | |
| Concomitant<br>Medications | X | | X | | X | X | X | X | |
| Physical Exam | X | | | | | | X | X | |
| Vital Signs | X | | X | | X | X | X | X | Height and weight will be assessed at screening; BP, pulse, respiration rate, and |

| | | | | | | | | | temperature will be assessed at each visit. Smoking status will be recorded at Screening |
|---|---|---|---|---|---|---|---|---|---|
| eDiary | X | X | X | X | X | X | X | X | Subjects will be provided eDiary to be completed at home daily and in-clinic. At home eDiary will include WI-NRS, AI-NRS, rescue medication, dose administration, and local skin tolerability. In clinic eDiary will include POEM and 5-D Pruritus Scale. eDiary will be reviewed at the baseline visit to determine eligibility. |
| POEM | X | | X | | X | X | X | X | Patient reported assessment by ePRO |
| 5-D Pruritus<br>Scale | X | | X | | X | X | X | X | Patient reported assessment by ePRO |
| IGA | X | | X | | X | X | X | X | Clinician assessment by eCOA |
| EASI | X | | X | | X | X | X | X | Clinician assessment by eCOA |
| Itch Numeric<br>Rating Scale<br>(NRS) | X | X | X | X | X | X | X | X | Patient reported assessment by ePRO |
| Clinical Labs | X | | | | | X | | X | Patients should fast for at least 8 hours before the test but optional at screening. Blood and urine for clinical |

| | | | | | | | | (if visit<br>occurs before<br>Day 28) | chemistry will be shipped to the central lab for processing. Chemistry, Hematology, Lipid Panel, and Urinalysis will be done at Screening and Day 28. Serology will only be done at Screening. Kits and lab manuals will be provided by a central lab. |
|---|---|---|---|---|---|---|---|---|---|
| Urine pregnancy test for WOCBP | X | | X | | | X | X | X | |
| IWRS | | | X | | | | | | |
| Investigational<br>Product<br>compliance | | | Х | | X | X | | X | Weights of dispensed and collected bottles to be recorded following instructions provided to sites. |
| Dispense study drug | | | X | | X | | | | |
| Application of study drug | | | X | X | X | X | | | First application of study drug will occur in the office under the supervision of the study staff. |
| Phone call to subjects | | X | | X | | | | | Call to initiate washout phase will be placed once results of screening clinical |

| | | | | | | | | | labs are finalized. Call on Day 5 will be made to counsel subjects on the use of IP and eDiary recordings, as well as answer any questions. |
|---|---|---|---|---|---|---|---|---|---|
| Collect study drug | | | | | X | X | | X | |
| Study counseling | X | X | X | X | X | X | | | Subjects will be counseled at each visit on the appropriate use of IP, eDiary entries and use. |
| AE monitoring | X | | X | | X | X | X | X | AE will be monitored from screening to follow-up. After informed consent, but prior to study drug administration, only SAEs caused by a protocolmandated intervention will be collected |

# **APPENDIX A continued:**

# **Schedule of eDiary and Efficacy Assessments**

eDiary (ePRO) is provided to subjects at the screening visit for daily entry at home (e.g., application on smartphone). Questionnaires and clinician assessments are recorded via ePRO/eCOA (e.g., tablet) or CRF during the site visits per schedule of events. Additional patient reported information include rescue medication use, dose administration confirmation, and adjunctive therapy use.

| Device | Assessment | Frequency and Duration of Assessment |
|---|---|---|
| eDiary | WI-NRS | Once daily from Screening visit through the Follow-up visit |
| eDiary | AI-NRS | Once daily from Screening visit through the Follow-up visit |
| eDiary | Local Tolerability | Once daily from Day 1 to Day 7 of treatment |
| eDiary | POEM | Patient reported at site visits |
| eDiary | 5-D Pruritus Scale | Patient reported at site visits |
| eCOA/CRF | IGA | Clinician assessment at site visits |
| eCOA/CRF | EASI | Clinician assessment at site visits |

# APPENDIX B: EXCLUDED MEDICATIONS/THERAPY

Excluded medication/therapy is listed below. The use of an excluded medication/therapy is a protocol violation and must be recorded in the CRF.

# Within 4 weeks prior to Baseline through the Follow-up period

- Systemic immunosuppressive/immunomodulating drugs (i.e., methotrexate, cyclosporine, etc.).
- Immunoglobulin or blood products.
- Systemic corticosteroids (oral, IV, injectable)
- NK1-R antagonists
- Class III or higher topical corticosteroids or any topical anti-pruritic therapies (other than stable doses of low- or mid-potency topical corticosteroids or bland emollients)
- Systemic therapies with recognized anti-pruritic (e.g. tricyclic antidepressants, sedatives, tranquilizers, gabapentin, marijuana or other cannabinoids, opioid receptor agonists/antagonists) or pruritic (e.g. opioids, angiotensin-converting enzyme inhibitors, cocaine, antimalarials) properties
  - Stable doses of oral H1 antihistamines will be permitted
- Systemic immunosuppressive/immunomodulatory therapies (including but not limited to PDE4 inhibitors, cyclosporine, mycophenolate-mofetil, methotrexate, azathioprine, interferon-gamma, or phototherapy)
- Allergen immunotherapy
- Any investigational therapy
- Strong CYP3A4 inhibitors, such as
  - boceprevir
  - clarithromycin
  - cobicistat
  - conivaptan
  - danoprevir and ritonavir
  - diltiazem
  - elvitegravir and ritonavir
  - regular grapefruit juice consumption
  - idelalisib
  - indinavir and ritonavir
  - itraconazole
  - ketoconazole
  - lopinavir and ritonavir
  - nefazodone
  - nelfinavir
  - paritaprevir and ritonavir and (ombitasvir and/or dasabuvir)
  - posaconazole
  - ritonavir

- saquinavir and ritonavir
- telaprevir
- tipranavir and ritonavir
- troleandomycin
- voriconazole

# Within 2 weeks prior to Baseline through the Follow-up period

- High-potency topical corticosteroids (Class 1-3). The use of low- to mid-potency topical corticosteroids (Class 4-7), inhaled corticosteroids, or intranasal corticosteroids will be allowed.
- Use of crisaborole ointment.
- Systemic antibiotics.
- Bleach baths or topical coal tar.
- Topical calcineurin inhibitor use (e.g., pimecrolimus, tacrolimus).
- New onset use of systemic antihistamines.
- UVA or UVB phototherapy
- Topical and oral antibiotics/antiviral/antifungal/antiseptic agents
- Topical probiotics
- Topical antihistamines.
- The use of intranasal and oral antihistamines will be allowed<sup>a</sup>.
- a Subjects following stable regimens (≥2 weeks consistent for intranasal and 3 months for oral use before study baseline) with systemic antihistamines are permitted to continue use but should not alter the dose or stop the regimen while in the study within 1 week prior to Baseline.

#### **Biologics**

- Cell-depleting agents, including but not limited to rituximab: within 6 months of baseline.
- Infliximab, adalimumab, golimumab, certolizumab pegol, abatacept, etanercept, anakinra, and dupilumab: within 12 weeks of baseline, or 5 half-lives, whichever is longer.
- Other biologics: within 12 weeks of Baseline, or 5 half-lives (if known), whichever is longer.

# APPENDIX C: EASI SCORE

#### How to Use EASI

The EASI scoring system uses a **defined process** to grade the **severity of the signs** of eczema and the **extent affected**:

### 1. Select a body region

Four body regions are considered separately:

- Head and neck
- · Trunk (including the genital area)
- Upper extremities
- · Lower Extremities (including the buttocks)

### 2. Assess the extent of eczema in that body region

Each body region has potentially 100% involvement. Using the table below, give each respective body region a score of between 0 and 6 based on the percentage involvement. Precise measurements are not required.

| % involvement | 0 | 1-9% | 10 - 29% | 30 - 49% | 50 - 69% | 70 - 89% | 90 - 100% |
|---|---|---|---|---|---|---|---|
| Region score | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

To aid in your body region grading you can use the diagrams in Appendix 1.

# Assess the severity of each of the four signs in that body region:

- 1. Erythema
- 2. Edema/papulation
- 3. Excoriation
- 4. Lichenification

Further explanations of these terms can be found in FAQ's (Appendix 4)

Grade the severity of each sign on a scale of 0 to 3:

| 0 | None |
|---|----------|
| 1 | Mild |
| 2 | Moderate |
| 3 | Severe |

- Take an average of the severity across the involved region.
- ✓ Half points may be used e.g. 2.5.
- ✓ Palpation may be useful in assessing edema/papulation as well as lichenification

To aid your severity grading, a photographic atlas of suggested categories is available in Appendix 2

Remember: Include only inflamed areas in your assessment; do not include xerosis (dryness), ichthyosis, keratosis pilaris, urticaria, infection (unless there is underlying eczema), or post inflammatory pigmentation changes.

EASI guidance December 14

# How to record your scores

The assessed parameters are inserted into a table (example shown below for age≥8 years). The final EASI score ranges from 0-72.

| Body region | Erythema | | Edema/<br>papulation | Excoriation | Lichenification | Area score | Multiplier | Score |
|---|---|---|---|---|---|---|---|---|
| Head/neck | ( | + | + | + | ) | x | x0.1 | |
| Trunk | ( | + | + | + | ) | x | × 0.3 | |
| Upper extremities | ( | + | + | + | ) | x | x 0.2 | |
| Lower extremities | ( | + | + | + | ) | x | x 0.4 | |
| The final EASI score is the sum of the 4 region scores | | | | | | | | |

Two forms of the EASI scoring system are available depending on the age of the patients. The multipliers for the region score are different in the under 8's version to reflect the relative proportion of body regions in young children:

- Patients 8 years or above
- Patients under 8 years of age.

The forms can be found in appendix 3.1 and 3.2 and also as word documents on the HOME website (www.homeforeczema.org)

# Score each region from 0 to 100%



EASI guidance December 14

Protocol PRB244-01

Amendment 3 28-FEB-2020
Appendix 2: Eczema Area and Severity Index (EASI) -lesion severity atlas



EASI guidance December 14

Protocol PRB244-01

## Appendix 3.1: Eczema Area and Severity Index (EASI) case report form – age <8 years

Area of Involvement: Each body region has potentially 100% involvement. Score <u>0 to 6</u> based on the following table:

| % | involvement | 0 | 1-9% | 10 - 29% | 30 - 49% | 50 - 69% | 70 - 89% | 90 - 100% |
|---|---|---|---|---|---|---|---|---|
| R | tegion score | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

Severity of Signs: Grade the severity of each sign on a scale of 0 to 3:

| 0 | None |
|---|----------|
| 1 | Mild |
| 2 | Moderate |
| 3 | Severe |

- ✓ Take an average of the severity across the involved area.
- ✓ Half points may be used e.g. 2.5.

#### Scoring table:

| | | thema<br>0-3) | Edema/<br>Papulation | Excoriation<br>(0-3) | Lichenification (0-3) | Region score<br>(0-6) | Multiplier | Score per body region |
|---|---|---|---|---|---|---|---|---|
| Body region | | | (0-3) | | | | | |
| Head/neck | ( | + | + | + | ) | x | X 0.2 | |
| Trunk | ( | + | + | + | ) | x | X 0.3 | |
| Upper extremities | ( | + | + | + | ) | x | X 0.2 | |
| Lower extremities | ( | + | + | + | ) | х | X 0.3 | |
| The final EASI score is the sum of the 4 region scores: | | | | | | | | |
| | | | | | | | | (0-72) |

## Appendix 3.2: Eczema Area and Severity Index (EASI) case report form - age≥8 years

<u>Area of Involvement:</u> Each body area has potentially 100% involvement. Score <u>0 to 6</u> based on the following table:

| % involvement | 0 | 1-9% | 10 - 29% | 30 - 49% | 50 - 69% | 70 - 89% | 90 - 100% |
|---|---|---|---|---|---|---|---|
| Region score | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

Severity of Signs: Grade the severity of each sign on a scale of 0 to 3:

| 0 | None |
|---|----------|
| 1 | Mild |
| 2 | Moderate |
| 3 | Severe |

- Take an average of the severity across the involved area.
- ✓ Half points may be used e.g. 2.5.

#### Scoring table:

| Body region | | :hema<br>)-3) | Edema/<br>Papulation<br>(0-3) | Excoriation<br>(0-3) | Lichenification(0-<br>3) | Region score<br>(0-6) | Multiplier | Score per body<br>region |
|---|---|---|---|---|---|---|---|---|
| Head/neck | ( | + | + | + | ) | x | X 0.1 | |
| Trunk | ( | + | + | + | ) | х | X 0.3 | |
| Upper extremities | ( | + | + | + | ) | x | X 0.2 | |
| Lower extremities | ( | + | + | + | ) | x | X 0.4 | |
| The final EASI score is the sum of the 4 region scores: | | | | | | | (0-72) | |

## Appendix 4 - Frequently Asked Questions

#### What is the difference between edema/papulation and lichenification?

Consider edema/papulation as corresponding to the acute signs of atopic dermatitis that reflect histological spongiosis. Lichenification are more firm thickened plaques with accentuation of the skin markings that develop as a result of prolonged scratching or rubbing in chronic disease. In darker skin types, follicular lichenification may present as firm flat-topped discrete papules. Grade these chronic lesions as lichenification.

#### How do I grade prurigo nodules?

Prurigo nodules are larger, deeper lesions as a result of chronic scratching and are graded as areas of lichenification.

#### How do I grade erythema in darker skin?

To avoid underestimating inflammation in patients with darker skin tones, take into account the underlying skin pigment when grading erythema. Often this means increasing your erythema grade by one level.

#### Can half-steps be used to assess lesion severity?

The original EASI validation study allowed for half steps. These may be helpful when trying to average the severity of a parameter over a region. For example, if there are some areas with an erythema grading of 2 and some areas more consistent with a severity of 3, 2.5 may be a good choice.

# What if most areas in a region are a severity grade of 1, but there are some areas that are a grade 3?

Attempt to average the severity across the involved areas in that region. If these areas are close to equal in size, a score of 2 would be most appropriate. If the majority of involved areas are a grade 1, a score of 1 or 1.5 is more appropriate. Be careful not to score the highest severity in a region but the average one.

#### How do I grade xerosis (dryness), ichthyosis and hyperlinear palms?

Unless there is active acute or chronic eczema overlying these findings, they are not included in the EASI assessment.

#### How precise should my assessment of eczema extent be?

The region scores, which reflect the extent of eczema, were designed and validated as rough estimates of the percentage of involved skin. Each region is given a score ranging from 0 to 6, based on a "ballpark" estimation of extent (see region score table in page 1). If you find it difficult to provide a rough estimate of disease extent, you can use the schematics in Appendix 1 to guide you. More time-consuming methods for evaluating disease extent such as the rule of nines or the 'palm' method are generally unnecessary, as the EASI was designed to be...easy.

# My patient has responded well to treatment and significantly improved since the last visit. Should I adjust the grading based on the patient's relative improvement?

No. The EASI is a static score, meaning that it is done independently at each time point to reflect current severity. You should grade the EASI per visit regardless of the previous status. Studies have shown that the EASI score has good responsiveness, meaning that overall it is sensitive to change and the improvement will be reflected in the total score.

#### Can the EASI be used in children?

Yes. The EASI is performed in the same method in all age groups, but the calculation of the final EASI score differs by age. When calculating the EASI, each of the 4 region scores is multiplied by a constant which reflects the relative contribution of that region to the total body surface area. For patients 8 years and older the multipliers are 0.1 for the head/neck, 0.2 for the upper extremities, 0.3 for the trunk and 0.4 for the lower extremities. Below 8 years of age the head/neck multiplier is increased to 0.2 while the lower extremities multiplier decreases to 0.3, consistent with the proportions of these regions in childhood. Refer to Appendix 3 for EASI forms by age.

# What happens if a child turns 8 during the course of the study? Which EASI formula should I use?

There are no clear-cut definitions for this situation. In general, if the study is a short term study such as an RCT lasting a few months — using the same formula throughout the trial is preferred, even if the child turns 8 during these months. Keeping the EASI formula consistent in this scenario can serve to preserve the EASI sensitivity to change (e.g. its change in response to treatment) without compromising the validity of the score.

In long term studies such as cohort studies lasting a year or longer, it is important to update the EASI formula based on the physical changes children go through. Switching to the age 8+ formula once a child is older is preferred in that scenario.

#### What do the terms erythema, edema/papulation, excoriation and lichenification mean?

These are key signs of atopic dermatitis. Recognizing and grading them properly requires training on the visual and physical exam consistent with these signs. Generally speaking, erythema is skin redness; edema/papulation refers to an elevation or swelling of the skin (that should be differed from lichenification below); excoriations are scratch marks that have broken the skin surface; and lichenification is a leathery thickening of the skin with exaggerated skin markings.

# APPENDIX D: PATIENT ORIENTED ECZEMA MEASURE (POEM)





| PC | EM for self-comple | tion | |
|---|---|---|---|
| | Dat | e: | |
| se for each of the<br>nable to answer. | e seven questions be | elow about your ec | zema. Please leave blank |
| now many days ha | s your skin been itch | ny because of your e | eczema? |
| 1-2 days | 3-4 days | 5-6 days | Every day |
| now many nights | has your sleep been | disturbed because o | of your eczema? |
| 1-2 days | 3-4 days | 5-6 days | Every day |
| now many days ha | s your skin been ble | eding because of yo | our eczema? |
| 1-2 days | 3-4 days | 5-6 days | Every day |
| now many days ha | s your skin been we | eping or oozing clea | ar fluid because of your |
| 1-2 days | 3-4 days | 5-6 days | Every day |
| now many days ha | s your skin been cra | cked because of you | ur eczema? |
| 1-2 days | 3-4 days | 5-6 days | Every day |
| now many days ha | s your skin been flak | ing off because of y | our eczema? |
| 1-2 days | 3-4 days | 5-6 days | Every day |
| now many days ha | s your skin felt dry o | r rough because of | your eczema? |
| 1-2 days | 3-4 days | 5-6 days | Every day |
| | Total POEM Sco | ore (Maximum 2 | 28): |
| | se for each of the<br>nable to answer.<br>now many days ha<br>1-2 days | Dates for each of the seven questions be nable to answer. In ow many days has your skin been itch 1-2 days 3-4 days now many days has your skin been ble 1-2 days 3-4 days now many days has your skin been were 1-2 days 3-4 days now many days has your skin been were 1-2 days 3-4 days now many days has your skin been craft 1-2 days 3-4 days now many days has your skin been flake 1-2 days 3-4 days now many days has your skin been flake 1-2 days 3-4 days now many days has your skin felt dry of 1-2 days 3-4 days | 1-2 days 3-4 days 5-6 days now many days has your sleep been disturbed because of 1-2 days 3-4 days 5-6 days now many nights has your sleep been disturbed because of 1-2 days 3-4 days 5-6 days now many days has your skin been bleeding because of you 1-2 days 3-4 days 5-6 days now many days has your skin been weeping or oozing cleat 1-2 days 3-4 days 5-6 days now many days has your skin been cracked because of you 1-2 days 3-4 days 5-6 days now many days has your skin been flaking off because of you 1-2 days 3-4 days 5-6 days now many days has your skin been flaking off because of you 1-2 days 3-4 days 5-6 days now many days has your skin felt dry or rough because of you 1-2 days 3-4 days 5-6 days |

© The University of Nottingham





#### POEM for self-completion

#### How is the scoring done?

Each of the seven questions carries equal weight and is scored from 0 to 4 as follows:

> No days = 0 1-2 days = 1 3-4 days = 2 5-6 days = 3 Every day = 4

#### Note:

- If one question is left unanswered this is scored 0 and the scores are summed and expressed as usual out of a maximum of 28
- If two or more questions are left unanswered the questionnaire is not scored
- If two or more response options are selected, the response option with the highest score should be recorded

#### What does a poem score mean?

To help patients and clinicians to understand their POEM scores, the following bandings have been established (see references below):

| • 0 to 2 | = Clear or almost clear |
|------------|-------------------------|
| • 3 to 7 | = Mild eczema |
| •8 to 16 | = Moderate eczema |
| • 17 to 24 | = Severe eczema |
| • 25 to 28 | = Very severe eczema |

## Do I need permission to use the scale?

Whilst the POEM scale is protected by copyright, it is freely available for use and can be downloaded from: <a href="https://www.nottingham.ac.uk/dermatology">www.nottingham.ac.uk/dermatology</a>.

We do however ask that you register your use of the POEM by e-mailing <a href="mailto:cebd@nottingham.ac.uk">cebd@nottingham.ac.uk</a> with details of how you would like to use the scale, and which countries the scale will be used in.

#### References

Charman CR, Venn AJ, Williams HC. The Patient-Oriented Eczema Measure: Development and Initial Validation of a New Tool for Measuring Atopic Eczema Severity From the Patients' Perspective. Arch Dermatol. 2004;140:1513-1519

Charman CR, Venn AJ, Ravenscroft JC, Williams HC. Translating Patient-Oriented Eczema Measure (POEM) scores into clinical practice by suggesting severity strata derived using anchor-based methods. Br J Dermatol. Dec 2013; 169(6): 1326–1332.

© The University of Nottingham. The Patient Oriented Eczema Measure (POEM) scale is free to use. Permission is granted to reproduce and/or redistribute this material in its entirety without modification. Any use which falls outside this remit requires the express consent of the copyright owner.

# **APPENDIX E: IGA**

| Score | Category | Definition |
|---|---|---|
| 0 | Clear | Minor residual discoloration, no erythema or induration/papulation, no oozing/crusting |
| 1 | Almost Clear | Trace faint pink erythema with almost no induration/papulation and no oozing/crusting |
| 2 | Mild Disease | Faint pink erythema with mild induration/papulation and no oozing/crusting |
| 3 | Moderate<br>Disease | Pink-red erythema with moderate induration/papulation and there may be some oozing/crusting |
| 4 | Severe Disease | Deep/bright red erythema with severe induration/papulation with oozing/crusting |

## **APPENDIX F: 5-D PRURITUS SCALE**

## 5-D Pruritus Scale

| 1. | <b>Duration</b> : D | uring the la | st 2 weeks, I | eeks, how many hours a day have you been itching? | | | |
|---|---|---|---|---|---|---|---|
| | Le | ess than 6hrs/o | day 6-12 hrs/c | day 12-18 h | rs/day 18-23 | hrs/day | All day |
| 2. | Degree: Ple | ase rate the | intensity of | your itching | g over the pa | st 2 weeks | |
| | | Not present | Mild | Mode: | rate Se | evere | Unbearable 5 |
| 3. | Direction: O | | st 2 weeks h | as your itch | ing gotten be | tter or wors | e compared to the |
| | | Completely resolved | Much better,<br>still preser | but Little bi | | hanged | Getting worse |
| 4. | Disability:<br>weeks | Rate the im | pact of your | itching on t | he following a | activities ove | er the last 2 |
| | Sleep | Never<br>affects sleep | Occasional<br>delays<br>falling aslee | dela | ently and occ<br>ys wake | alling asleep<br>casionally<br>es me up<br>night | Delays falling asleep and frequently wakes me up at night |
| | | N/A | Never<br>affects<br>this activity | Rarely<br>affects<br>this activity | Occasionally<br>affects<br>this activity | Frequently<br>affects<br>this activity | affects |
| | Leisure/Soci | al 🗌 | $\Box$ | | | | |
| | Housework/<br>Errands | | | 2 | 3 | 4 | 5 |
| | Work/School | | | 2 | 3 | 4 | 5 |
| 5. | | t 2 weeks. I<br>y. | f a body part | | resent in the<br>d, choose the | one that is | arts of your body closest |
| | Head/Scalp<br>Face<br>Chest<br>Abdomen<br>Back<br>Buttocks<br>Thighs<br>Lower legs | | Forea Upper Points | of Hands/Fi<br>rms<br>r Arms<br>s of Contact<br>waistband, i | ingers<br>w/ Clothing<br>undergarmen | Present | |

## APPENDIX G: PATIENT REPORTED LOCAL TOLERABILITY

PATIENT ASSESSMENT OF LOCAL SKIN TOLERABILITY AT APPLICATION SITE(S)

SUBJECT AGE RANGE: 12 years old and above

## **INSTRUCTIONS:**

Please examine all of your skin lesions that are treated with B244 topical solution. Please circle one score for each category that best describes the changes you observed in all skin lesions. For each day of the first 7 days of treatment, please examine all skin lesions at approximately the same time every day.

| DAY OF TREATMENT | (1-7): |
|------------------|----------|
| TIME OF DAY: | AM or PM |

| | SKIN REDNESS AND/OR COLOR CHANGE AT APPLICATION SITE | |
|---|---|---|
| Score | Grade | Definition |
| 0 | None | No new redness or new color change; no new increase in redness or new increase in color change |
| 1 | Mild | Slight increase in redness or slight increase in color change |
| 2 | Moderate | Increase in redness or increase in color change |
| 3 | Severe | Intense redness or intense color change |

| | ITCHING AT APPLICATION SITE | |
|---|---|---|
| Score | Grade | Definition |
| 0 | None | No new itching or new scratching |
| 1 | Mild | Slight increase in itching or slight increase in scratching |
| 2 | Moderate | Increase in itching or increase in scratching that is not disturbing sleep |
| 3 | Severe | Increase in itching or increase in scratching that is disturbing sleep |

| BURNING AND/OR STINGING AT APPLICATION SITE | | |
|---|---|---|
| Score | Grade | Definition |
| 0 | None | No new burning or new stinging |
| 1 | Mild | Slight increase in warm or tingling sensation that is not bothersome |
| 2 | Moderate | Increase in warm or tingling sensation that is bothersome |
| 3 | Severe | Hot or stinging sensation that is causing definite discomfort |

| | PAIN AND/OR TENDERNESS AT APPLICATION SITE | |
|---|---|---|
| Score | Grade | Definition |
| 0 | None | No new pain or new tenderness |
| 1 | Mild | Slight increase in pain or slight increase in tenderness that is not bothersome |
| 2 | Moderate | Increase in pain or increase in tenderness that is bothersome |
| 3 | Severe | Intense pain or intense tenderness causing definite discomfort or disturbing sleep |

| NEW OR CHANGING RASH AT APPLICATION SITE | | |
|---|---|---|
| Score | Grade | Definition |
| 0 | None | No new rash or no change in rash (such as swelling, fullness, or blistering) |
| 1 | Mild | Slight new rash or slight increase in rash (such as swelling, fullness, or blistering) that is not bothersome |
| 2 | Moderate | New rash or increase in rash (such as swelling, fullness, or blistering) that is bothersome |
| 3 | Severe | Significant new rash or significant increase in rash (swelling, fullness, or blistering) causing discomfort |